

## **SPONSOR:**

Comprehensive Cancer Trial Centre (CCTU), Department of Clinical Oncology, The Chinese University of Hong Kong

## TITLE:

An open-label phase II study of pembrolizumab in East Asian patients with advanced/metastatic acral lentiginous melanoma

### IND NUMBER:

**EudraCT NUMBER (Studies in Europe only):** 



# **Version Updates:**

| Version | Date | Details of Update | Page | Notes/References |
|---------|---------|-----------------------------|-------|------------------|
| 1.1 | 16-Jun- | Addition of Table 6.2 – | 32-33 | |
| | 2016 | describes 'Second-course | ļ | |
| | | phase [Retreatment with | | |
| | | pembrolizumab]' | | |
| | | Table 9.1 – Only 100mg/4ml | 55 | |
| | | pembrolizumab vials will be | | |
| | | supplied for this study by | | |
| | | Merck | | |

| Version | Date | Details of Update | Page | Notes/References |
|---|---|---|---|---|
| 1.2 | 9-Oct-2018 | Addition of Table 8 — describes 'Modification and Toxicity Management Guildlines for Immunerelated AEs Associated with pembrolizumab' | 55-57 | |



## 1.0 TRIAL SUMMARY

| Abbreviated Title | Pembrolizumab in advanced/metastatic acral lentiginous melanoma |
|---|---|
| Trial Phase | П |
| Clinical Indication | Malignant melanoma – acral lentiginous type, palliative intent |
| Trial Type | Clinical |
| Type of control | Single-arm phase II Simon Minimax Design |
| Route of administration | IV |
| Trial Blinding | Open-label |
| Treatment Groups | Single-arm |
| Number of trial subjects | 28 |
| Estimated enrollment period | July 2016 June 2019 |
| Estimated duration of trial | 24 months enrollment, duration of trial 42 months |
| Duration of Participation | 42 months |

## 2.0 TRIAL DESIGN

## 2.1 Trial Design

A single-arm, open-label phase II clinical trial of pembrolizumab at 200mg IV infusion every 3 weeks in patients with metastatic/inoperable advanced acral lentiginous melanoma.



### 2.2 Trial Diagram



### 3.0 OBJECTIVE(S) & HYPOTHESIS(ES)

#### 3.1 Primary Objective(s) & Hypothesis(es)

### **Objective:**

To determine the Overall Response Rate (ORR), as defined as rate of complete response (CR) and partial response (PR) as per RECIST 1.1 in biological treatment-naïve patients with acral lentiginous melanoma treated with pembrolizumab

### Hypothesis:

Given the differing biology of acral lentiginous melanoma, we hypothesize that patients with acral lentiginous melanoma may have a different ORR as reported in prior studies with pembrolizumab in the Western population, of which the superficial spreading subtype is the majority. This may be attributable to the fact that the molecular genomic landscape of acral lentiginous melanoma is different from superficial spreading melanoma with higher incidence of c-KIT and lower incidence of BRAF mutations, we would expect the duration of treatment response may possibly be different as these factors have potential impact on treatment resistance pathways. There have been no large-scale studies documenting the



pharmacokinetics of pembrolizumab in East Asians, and we believe that there may possibly be distinct differences given differing body habitus.

### 3.2 Secondary Objectives

- 1. Assessment of response duration (time from best overall response of PR or CR to time of first documented disease progression)
- 2. Determine the Clinical Benefit Rate (CBR) of pembrolizumab treatment naïve acral lentiginous melanoma patients as defined by rate of CR + PR and stable disease (SD) of >/= 6 months
- 3. Progression-free survival (PFS)
- 4. Overall survival (OS)
- 5. Response assessment as per the Immune-related Response Criteria (irRC) and its correlation with survival
- 6. Continual assessment of adverse events as per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 4.0).

## 3.3 Exploratory Objectives

- 1. Incidence of baseline PD-L1 expression in acral lentiginous melanoma in East Asians and its potential prognostic and predictive implications
- 2. Effects of pembrolizumab on PD-L1 expression as assessed by on-treatment biopsies and its potential prognostic and predictive implications
- 3. Pharmacokinetic assessments in the East Asian population -- Peak and trough blood samples to be obtained and pembrolizumab serum concentrations to be quantified with a validated electrochemiluminsecent assay

## 4.0 BACKGROUND & RATIONALE

### 4.1 Background

Refer to the Investigator's Brochure (IB)/approved labeling for detailed background information on MK-3475.

## 4.1.1 Pharmaceutical and Therapeutic Background

The importance of intact immune surveillance in controlling outgrowth of neoplastic transformation has been known for decades. Accumulating evidence shows a correlation between tumor-infiltrating lymphocytes (TILs) in cancer tissue and favorable prognosis in various malignancies. In particular, the presence of CD8+ T-cells and the ratio of CD8+



effector T-cells / FoxP3+ regulatory T-cells seems to correlate with improved prognosis and long-term survival in many solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. The normal function of PD-1, expressed on the cell surface of activated Tcells under healthy conditions, is to down-modulate unwanted or excessive immune responses, including autoimmune reactions. PD-1 (encoded by the gene Pdcd1) is an Ig superfamily member related to CD28 and CTLA-4, which has been shown to negatively regulate antigen receptor signaling upon engagement of its ligands (PD-L1 and/or PD-L2). The structure of murine PD-1 has been resolved. PD-1 and family members are type I transmembrane glycoproteins containing an Ig Variable-type (V-type) domain responsible for ligand binding and a cytoplasmic tail which is responsible for the binding of signaling The cytoplasmic tail of PD-1 contains 2 tyrosine-based signaling motifs, an immunoreceptor tyrosine-based inhibition motif (ITIM) and an immunoreceptor tyrosine-Following T-cell stimulation, PD-1 recruits the tyrosine based switch motif (ITSM). phosphatases SHP-1 and SHP-2 to the ITSM motif within its cytoplasmic tail, leading to the dephosphorylation of effector molecules such as CD3ζ, PKCθ and ZAP70 which are involved in the CD3 T-cell signaling cascade. The mechanism by which PD-1 down modulates T-cell responses is similar to, but distinct from that of CTLA-4 as both molecules regulate an overlapping set of signaling proteins. PD-1 was shown to be expressed on activated lymphocytes including peripheral CD4+ and CD8+ T-cells, B-cells, T regs and Natural Killer cells. Expression has also been shown during thymic development on CD4-CD8- (double negative) T-cells as well as subsets of macrophages and dendritic cells. The ligands for PD-1 (PD-L1 and PD-L2) are constitutively expressed or can be induced in a variety of cell types, including non-hematopoietic tissues as well as in various tumors. Both ligands are type I transmembrane receptors containing both IgV- and IgC-like domains in the extracellular region and contain short cytoplasmic regions with no known signaling motifs. Binding of either PD-1 ligand to PD-1 inhibits T-cell activation triggered through the T-cell receptor. PD-L1 is expressed at low levels on various non-hematopoietic tissues, most notably on vascular endothelium, whereas PD-L2 protein is only detectably expressed on antigen-presenting cells found in lymphoid tissue or chronic inflammatory environments. PD-L2 is thought to control immune T-cell activation in lymphoid organs, whereas PD-L1 serves to dampen unwarranted T-cell function in peripheral tissues. Although healthy organs express little (if any) PD-L1, a variety of cancers were demonstrated to express abundant levels of this T-cell inhibitor. PD-1 has been suggested to regulate tumor-specific T-cell expansion in subjects with melanoma (MEL). This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention.

Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. Keytruda<sup>TM</sup> (pembrolizumab) has recently been approved in the United Stated for the treatment of patients with unresectable or metastatic melanoma and



disease progression following ipilumumab and, if BRAF V600 mutation positive, a BRAF inhibitor.

#### 4.1.2 Preclinical and Clinical Trial Data

Refer to the Investigator's Brochure for Preclinical and Clinical data.

#### 4.2 Rationale

### 4.2.1 Rationale for the Trial and Selected Subject Population

Whilst there is a low incidence of melanoma reported in East Asian regions (< 1 per 100,000) including China, Taiwan, Hong Kong and Singapore, the most common subtype in these regions has been reported as cutaneous acral lentiginous melanoma, which comprises approximately 50-58% in reported series[1]. This is in contrast to only 2% to 3% reported in Western populations. Conversely, the typical superficial spreading melanomas found that account for approximately 50-70% of melanomas in the Western population is less common in East Asia (5% - 37%). Acral lentiginous melanomas are usually present in areas with little to no sun exposure such as palms, soles and nail apparatus, which is thought to be UVprotected by the thickened stratum corneum and the nail matrix. The aetiology of acral melanoma in Asia remains to be determined, although observational studies have suggested that repeated trauma to the hands and feet, the exposure to agricultural chemicals[2] as well as more physically pressured sites (such as center area of heels and inner forefoot) may be contributory factors to their development[3]. Acral melanomas harbour a higher rate of genomic amplifications than other cutaneous melanomas. BRAF and RAS mutations are less common, whilst a higher incidence of KIT mutations have been reported[4, 5]. Studies have established acral melanoma as distinct from common cutaneous melanoma at the genomic level, with copy number profiling revealing a higher degree of aneuploidy in acral and mucosal than cutaneous melanoma[4]. Recently, the pattern of somatic alterations in acral melanoma was identified[6, 7], suggesting that in addition to point mutations, acral melanoma drivers are also activated by large-scale genomic rearrangements.

The distinct mechanism of action of anti-programmed-death-receptor-1 (PD-1) antibodies, which increase tumour cell killing peripherally by cytotoxic T lymphocytes, has recently been shown to have activity in patients with ipilimumab refractory melanoma[8]. Immune checkpoint inhibitors have exhibited unusual kinetics of response, with slow responses in some patients on-going for a year or more, late responses at 6-12 months, and unprecedented progression followed by regression in a significant proportion of patients. Similar observations of pseudo-progression have also been noted with the PD-1 antibody nivolumab, in both melanoma and in non-small cell lung cancer[9]. This phenomenon has been attributed to delayed immune activity and subsequent oedema.

Pembrolizumab (MK-3475), a highly selective humanized monoclonal IgG4-kappa isotype antibody against PD-1 has been shown to have potent anti-tumour activity at different doses and schedules in patients with melanoma. Results of the open-label, expansion cohort of the



KEYNOTE-001 multi-centre trial consisting of over 170 patients with advanced melanoma that progressed after at least two ipilimumab doses have recently been published showing an overall response rate (ORR) of 26% in both the 10mg/kg Q3W and 2mg/kg Q3W schedules studied[10]. The treatment was well tolerated with similar safety profiles in both treatment groups. There were no treatment related deaths. Common drug-related adverse events were those expected of this particular class of agents, with fatigue, pruritis and skin rash being most common. Specifically, this international multi-centre trial was conducted in Australia, Canada, France and the USA and the demographics of patients in this study were predominantly White Caucasians (97%). There were only 3 Asian patients (2%) in the entire trial. From published results, there is no mention on the distribution of melanoma subtypes in these patients. Presumably, the geographical location of where this study was conducted and the ethnicity of the patients recruited mean that the majority of patients suffered from superficial spreading melanoma and patients with acral lentiginous melanoma only formed a minority and may not have been adequately represented. Given the differing aetiological and pathogenomic factors between subtypes of malignant melanomas, whether the results obtained from prior international trials are applicable to patients with acral lentiginous melanoma, which is by far more common in the East Asian population, are called into question. In addition, there has been observation that patients whose tumour initially showed radiological progression have subsequently proven to yield benefit in terms of clainical and radiological assessment. The underlying mechanism of such observation is unknown.

In Hong Kong, the treatment of metastatic melanoma is also challenged by limited therapeutic options. At present, ipilimumab has yet to obtain approval from the Department of Health in the Hong Kong Special Administrative Region (HKSAR). Beyond conventional cytotoxics, vemurafenib is the only targeted agent registered in the HKSAR for malignant melanomas carrying a BRAF V600E mutation. However, the agent is currently not available within the government reimbursement program. As a result, the standard of care for most patients in our locality suffering from metastatic melanoma is conventional cytotoxics.

We believe it is prudent to assess the activity of pembrolizumab in a specific phase II trial in patients suffering from acral lentiginous melanoma in East Asia. Also, there appears to be a paucity of data on the pharmacokinetic properties of pembrolizumab in East Asians available in published literature. Given the fact that there is a difference in the average body habitus between East Asians and in Caucasians and Black/African-American ethnicities, this study will provide a good opportunity to study the pharmacokinetic profiles of pembrolizumab in the East Asian population.

#### 4.2.2 Rationale for Dose Selection/Regimen/Modification

An open-label Phase I trial (Protocol 001) is being conducted to evaluate the safety and clinical activity of single agent MK-3475. The dose escalation portion of this trial evaluated three dose levels, 1 mg/kg, 3 mg/kg, and 10 mg/kg, administered every 2 weeks (Q2W) in



subjects with advanced solid tumors. All three dose levels were well tolerated and no dose-limiting toxicities were observed. This first in human study of MK-3475 showed evidence of target engagement and objective evidence of tumor size reduction at all dose levels (1 mg/kg, 3 mg/kg and 10 mg/kg Q2W). No MTD has been identified to date. 10.0 mg/kg Q2W, the highest dose tested in PN001, will be the dose and schedule utilized in Cohorts A, B, C and D of this protocol to test for initial tumor activity. Recent data from other clinical studies within the MK-3475 program has shown that a lower dose of MK-3475 and a less frequent schedule may be sufficient for target engagement and clinical activity.

PK data analysis of MK-3475 administered Q2W and Q3W showed slow systemic clearance, limited volume of distribution, and a long half-life (refer to IB). Pharmacodynamic data (IL-2 release assay) suggested that peripheral target engagement is durable (>21 days). This early PK and pharmacodynamic data provides scientific rationale for testing a Q2W and Q3W dosing schedule.

A population pharmacokinetic analysis has been performed using serum concentration time data from 476 patients. Within the resulting population PK model, clearance and volume parameters of MK-3475 were found to be dependent on body weight. The relationship between clearance and body weight, with an allometric exponent of 0.59, is within the range observed for other antibodies and would support both body weight normalized dosing or a fixed dose across all body weights. MK-3475 has been found to have a wide therapeutic range based on the melanoma indication. The differences in exposure for a 200 mg fixed dose regimen relative to a 2 mg/kg Q3W body weight based regimen are anticipated to remain well within the established exposure margins of 0.5 – 5.0 for MK-3475 in the melanoma indication. The exposure margins are based on the notion of similar efficacy and safety in melanoma at 10 mg/kg Q3W vs. the proposed dose regimen of 2 mg/kg Q3W (i.e. 5-fold higher dose and exposure). The population PK evaluation revealed that there was no significant impact of tumor burden on exposure. In addition, exposure was similar between the NSCLC and melanoma indications. Therefore, there are no anticipated changes in exposure between different indication settings.

The rationale for further exploration of 2 mg/kg and comparable doses of pembrolizumab in solid tumors is based on: 1) similar efficacy and safety of pembrolizumab when dosed at either 2 mg/kg or 10 mg/kg Q3W in melanoma patients, 2) the flat exposure-response relationships of pembrolizumab for both efficacy and safety in the dose ranges of 2 mg/kg Q3W to 10 mg/kg Q3W, 3) the lack of effect of tumor burden or indication on distribution behavior of pembrolizumab (as assessed by the population PK model) and 4) the assumption that the dynamics of pembrolizumab target engagement will not vary meaningfully with tumor type.

The choice of the 200 mg Q3W as an appropriate dose for the switch to fixed dosing is based on simulations performed using the population PK model of pembrolizumab showing that the fixed dose of 200 mg every 3 weeks will provide exposures that 1) are optimally consistent with those obtained with the 2 mg/kg dose every 3 weeks, 2) will maintain individual patient



exposures in the exposure range established in melanoma as associated with maximal efficacy response and 3) will maintain individual patients exposure in the exposure range established in melanoma that are well tolerated and safe.

A fixed dose regimen will simplify the dosing regimen to be more convenient for physicians and to reduce potential for dosing errors. A fixed dosing scheme will also reduce complexity in the logistical chain at treatment facilities and reduce wastage.

#### 4.2.3 Rationale for Endpoints

#### 4.2.3.1 Efficacy Endpoints

The study shall be powered to determine its primary endpoint of establishing the ORR as defined as the rate of CR and PR as per RECIST 1.1 in biological treatment-naïve patients with acral lentiginous melanoma being treated with pembrolizumab. This is a suitable endpoint given the overall rarity of the disease, as ORR requires a smaller population to establish and can be compared with historical data of prior treatment regimens. The efficacy of treatment can also be attributed directly to the treatment itself, and not to the natural history of the disease.

Secondary endpoints of response and efficacy include 1) assessment of response duration, 2) CBR, 3) PFS, 4) OS as described in section 3.2.

Additional explorative assessment of response as per irRC and its correlation with survival will further add to the volume of data generated in various trials with checkpoint inhibitors, allowing investigators to better understand the notion of "immune response", and how that may be similar or different from traditional response assessments as determined by RECIST. Safety assessments and documented as per CTCAE 4.0 will be carried out throughout the duration of the study.

## 4.2.3.2 Biomarker Research

- 1. The incidence of PD-L1 expression in acral lentiginous melanoma in East Asians and its potential prognostic and predictive implications will be determined, as documented by the initial tumour specimen either from archival sample or a new biopsy. The genomic mutational landscape of acral melanomas in the East Asian population will be explored.
- 2. With the mandatory on-treatment biopsy, changes in PD-L1 expression (if any) after 2 doses of pembrolizumab can be assessed. Whether changes in PD-L1 expression in this situation may have a predictive or prognostic significance to pembrolizumab treatment will be explored.



3. Pharmacokinetics assessments of pembrolizumab in an East Asian population will be performed.

#### 5.0 METHODOLOGY

### 5.1 Entry Criteria

### 5.1.1 Diagnosis/Condition for Entry into the Trial

Diagnosis of histologically proven acral lentiginous melanoma with metastatic disease and/or not amenable to curative resection. Prior treatment with conventional cytotoxics (including, but not limited to DTIC, temozolomide, paclitaxel and carboplatin) is allowed. Prior treatment with ipilimumab (CTLA-4 inhibitor) is also allowed.

### 5.1.2 Subject Inclusion Criteria

In order to be eligible for participation in this trial, the subject must:

- 1. Be willing and able to provide written informed consent/assent for the trial.
- 2. Be  $\geq$  18 years of age on day of signing informed consent.
- 3. Have measurable disease based on RECIST 1.1.
- 4. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
- 5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
- 6. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

Table 1 Adequate Organ Function Laboratory Values

| System | Laboratory Value |
|------------------------------|-----------------------------------------------|
| Hematological | |
| Absolute neutrophil co (ANC) | ount ≥1,500 /mcL |
| Platelets | ≥100,000 / mcL |
| Hemoglobin | ≥9 g/dL or ≥5.6 mmol/L without transfusion or |



| | EPO dependency (within 7 days of assessment) |
|---|---|
| Renal | |
| Serum creatinine OR | ≤1.5 X upper limit of normal (ULN) <u>OR</u> |
| Measured or calculated <sup>a</sup> | |
| creatinine clearance | ≥60 mL/min for subject with creatinine levels > |
| (GFR can also be used in place | 1.5 X institutional ULN |
| of creatinine or CrCl) | |
| Hepatic | |
| Serum total bilirubin | ≤ 1.5 X ULN <u>OR</u> |
| | Direct bilirubin ≤ ULN for subjects with total |
| | bilirubin levels > 1.5 ULN |
| AST (SGOT) and ALT (SGPT) | ≤ 2.5 X ULN <u><b>OR</b></u> |
| AST (SOOT) and ALT (SOFT) | ≤ 5 X ULN for subjects with liver metastases |
| Albumin | $\geq$ 2.5 mg/dL |
| Coagulation | |
| | ≤1.5 X ULN unless subject is receiving |
| International Normalized Ratio | anticoagulant therapy |
| (INR) or Prothrombin Time | as long as PT or PTT is within therapeutic range |
| (PT) | of intended use of anticoagulants |
| | ≤1.5 X ULN unless subject is receiving |
| Activated Partial | anticoagulant therapy |
| Thromboplastin Time (aPTT) | as long as PT or PTT is within therapeutic range |
| | of intended use of anticoagulants |
| <sup>a</sup> Creatinine clearance should be | calculated per institutional standard. |

- 7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
- 8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
- 9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

### 5.1.3 Subject Exclusion Criteria

The subject must be excluded from participating in the trial if the subject:



- 1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapyor used an investigational device within 4 weeks of the first dose of treatment.
- 2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
- 3. Has a known history of active TB (Bacillus Tuberculosis)
- 4. Hypersensitivity to pembrolizumab or any of its excipients.
- 5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
- 6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
  - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
- 7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
- 8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least eight weeks prior to the first dose of trial treatment), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
- 9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.



- 10. Has known history of, or any evidence of active, non-infectious pneumonitis.
- 11. Has an active infection requiring systemic therapy.
- 12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
- 15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
- 16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
- 17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
- 18. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

#### 5.2 Baseline Procedures

#### 5.2.1 Baseline Clinical Assessment

Potential subjects will screened at a clinical visit, with specific clinical status requirements as per the criteria set above.

### 5.2.2 Baseline Imaging

Subjects who fulfill the above eligibility/exclusion criteria are to proceed with baseline contrast CT Brain, Thorax, Abdomen and Pelvis as baseline imaging assessment. Patients with brain metastases, provided that they have been i) treated, ii) radiologically proven to be stable for at least 8 weeks and iii) not on steroids, are allowed in the study.



## 5.2.3 Baseline Laboratory Investigations

Baseline laboratory investigations as specified above, including hepatitis and HIV screening shall be performed during the screening period.

## 5.2.4 Archival Tissue Sample or Fresh Biopsy

To be eligible for the study, subjects are required to have either:

i) Archival tissue available for correlative studies, with no interval treatment between the sample date and start of the study

Or

ii) Agreeable for a fresh biopsy at baseline prior to start of pembrolizumab dosing, if the above is not available.

#### 5.3 Trial Treatments

The treatment to be used in this trial is outlined below in Table 2

**Table 2 Trial Treatment** 

| Drug | Dose | Dose | Route of | Regimen/Treat | Use |
|---|---|---|---|---|---|
| | | Frequenc | Administr | ment Period | |
| | | у | ation | } | |
| Pembrolizumab | 200 mg | Q3W | IV<br>infusion | Day 1 of each 3 week cycle | Experimental |

Trial treatment should begin on the day of randomization or as close as possible to the date on which treatment is allocated/assigned.

#### 5.3.1 Dose Selection/Modification

## 5.3.1.1 Dose Selection

The rationale for selection of doses to be used in this trial is provided in Section 4.0 – Background and Rationale.



Details on preparation and administration of pembrolizumab (MK-3475) are provided in the Pharmacy Manual.

### 5.3.1.2 Dose Modification

Adverse events (both non-serious and serious) associated with pembrolizumab exposure may represent an immunologic etiology. These adverse events may occur shortly after the first dose or several months after the last dose of treatment. Pembrolizumab must be withheld for drug-related toxicities and severe or life-threatening AEs as per Table 3 below. See Section 5.6.1 and Events of Clinical Interest Guidance Document for supportive care guidelines, including use of corticosteroids.

Table 3

Dose Modification Guidelines for Drug-Related Adverse Events

| Toxicity | Hold<br>Treatm<br>ent For<br>Grade | Timing for Restarting<br>Treatment | Discontinue Subject |
|---|---|---|---|
| Diarrhea/Col<br>itis | 2-3 | Toxicity resolves to Grade 0-1. | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |
| AST, ALT, or Increased | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose. |
| Bilirubin | 3-4 | Permanently discontinue (see exception below) <sup>1</sup> | Permanently discontinue |
| Type 1<br>diabetes<br>mellitus (if<br>new onset) or<br>Hyperglycem<br>ia | T1DM<br>or<br>3-4 | Hold pembrolizumab for new onset Type 1 diabetes mellitus or Grade 3-4 hyperglycemia associated with evidence of beta cell failure. | Resume pembrolizumab when patients are clinically and metabolically stable. |
| Hypophysitis | 2-3 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |



| Toxicity | Hold<br>Treatm<br>ent For<br>Grade | Timing for Restarting<br>Treatment | Discontinue Subject |
|---|---|---|---|
| Hyperthyroid ism | 3 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |
| Hypothyroidi<br>sm | 2-4 | Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted | Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted. |
| Infusion<br>Reaction | 3-4 | Permanently discontinue | Permanently discontinue |
| Pneumonitis | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 3-4 | Permanently discontinue | Permanently discontinue |
| Renal Failure<br>or Nephritis | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 3-4 | Permanently discontinue | Permanently discontinue |
| All Other<br>Drug-Related<br>Toxicity <sup>2</sup> | 3 or<br>Severe | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |

Note: Permanently discontinue for any severe or Grade 3 drug-related AE that recurs or any life-threatening event.

<sup>1</sup> For patients with liver metastasis who begin treatment with Grade 2 AST or ALT, if AST or ALT increases by greater than or equal to 50% relative to baseline and lasts for at least 1 week then patients should be discontinued.

<sup>2</sup> Patients with intolerable or persistent Grade 2 drug-related AE may hold study medication at physician discretion. Permanently discontinue study drug for persistent Grade 2 adverse reactions for which treatment with study drug has been held, that do not recover to Grade 0-1 within 12 weeks of the last dose.



Dosing interruptions are permitted in the case of medical / surgical events or logistical reasons not related to study therapy (e.g., elective surgery, unrelated medical events, patient vacation, and/or holidays). Subjects should be placed back on study therapy within 3 weeks of the scheduled interruption, unless otherwise discussed with the Sponsor. The reason for interruption should be documented in the patient's study record.

### 5.3.2 Timing of Dose Administration

Trial treatment should be administered on Day 1 of each cycle after all procedures/assessments have been completed as detailed on the Trial Flow Chart (Section 6.0). Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial treatments will be administered on an outpatient basis.

Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

The Pharmacy Manual contains specific instructions for the preparation of the pembrolizumab infusion fluid and administration of infusion solution.

### 5.3.3 Trial Blinding/Masking

This is an open-label trial; therefore, the Sponsor, investigator and subject will know the treatment administered.

#### 5.3.4 Pharmacokinetics Assessment of Pembrolizumab

Previous investigations of pembrolizumab in patients who received doses of 1 to 10mg/kg every 2 weeks or 2 to 10mg/kg every 3 weeks have established steady state concentrations of pembrolizumab is reached by 18 weeks (~ 6 cycles) of repeated dosing with an every 3-week regimen.

To specifically explore pharmacokinetic properties of pembrolizumab in an East Asian population, the following pharmacokinetic sampling plan has been incorporated into this study

Pharmacokinetic samples are to be drawn at the following time-points:



| Study Day | Time (Event hours) | Time (Relative to dosing) (hr:min) |
|---|---|---|
| CIDI | 0 hrs (pre-dosing) | 00:00 |
| C1D1 | 30 mins (End-of-infusion) | 00:30 |
| C1D1 | 3 hrs (post infusion) | 03:00 |
| C1D2 | | 24:00 to 36:00 |
| C1D8 | | 168:00 |
| C2D1 | 0 (pre-dosing) | 00:00 |
| C6D1 (steady state) | 0 (pre-dosing) | 00:00 |

Blood samples should be drawn from a site other than the infusion site (ie, contralateral arm) on days of infusion. All samples collected pre-dose should be taken just prior to the administration, and end-of-infusion (EOI) samples should be taken as close to EOI as possible (preferably 2 minutes prior to EOI) on the contralateral arm (ie, the arm not for the infusion). If the infusion was interrupted, the reason for interruption should also be documented on the CRF. Blood samples will be processed to collect serum. The serum samples will be analyzed by an ELISA method. Further details of blood collection, labeling, processing, storage can be found in the procedure manual.

### 5.3.5 On-Treatment Biopsy

On-treatment biopsy shall be performed if deemed safe by the investigators and technically feasible. Preferably, the on-treatment biopsy shall be of the same lesion that prior tissue was obtained from (either archival or fresh sample), shall be performed at 6 weeks (after 2 doses of pembrolizumab) after start of study treatment, before the 3<sup>rd</sup> dose of pembrolizumab.

#### 5.3.6 On-Treatment Radiological Assessments

Response assessments with CT imaging shall be performed every 6 weeks (2 cycles of pembrolizumab) in the first 24 months, then every 9 weeks (3 cycles of pembrolizumab) should the subject continues on study.

### 5.3.7 Continuation of Treatment Beyond RECIST Progression

For subjects who have been determined to have progressive disease as per RECIST, but who may appear to be benefiting from treatment, may continue with pembrolizumab at the



investigators' discretion. Mandatory reassessment imaging must be performed with a time interval of at least 4 weeks after the latest imaging. Should there be further evidence of disease progression, further treatment shall be discontinued. The time of disease progression shall be dated back to the time of the prior imaging.

Subjects shall be followed beyond disease progression and discontinuation from study. Further lines of treatment (if any) received by the subjects shall be documented. Survival data shall be obtained.

#### 5.4 Treatment Allocation and Statistical Considerations

This is an open-label single-arm phase II study. There is no randomization of patients. All patients will receive the investigational product.

The primary objective is to determine the ORR (CR+PR) of pembrolizumab in patients with acral lentiginous melanoma who have not received prior anti-PD-1 or anti-PD-L1 treatment. Based on literature review, the ORR of first line treatment with checkpoint inhibitors of melanoma in general is in the range of 32-40%.

We assume that the ORR achievable with pembrolizumab in acral lentiginous melanoma would be similar.

The Simon's Minimax two-stage phase II design was used to calculate sample size. We consider the pembrolizumab to be inactive if the treatment response rate (confirmed CR and PR) is  $\leq 10\%$ , and consider the pembrolizumab as active if the treatment response rate is  $\geq 30\%$ . Therefore, assuming  $P_0 = 0.10$ ,  $P_1 = 0.30$ , and the type I error of 0.05 with power of 80%, the sample size and stopping rule are as follow:

<u>Stage I:</u> Accrue 15 patients; if 1 or less of the 15 patients are non-responders, we would stop the study and conclude pembrolizumab as inactive, otherwise proceed to stage II.

<u>Stage II:</u> Accrue an additional 10 patients. If 5 or less of the 25 patients are non-responders, pembrolizumab will be deemed inactive.

Using this phase II design the average sample size is 19.5 patients if the treatment is in fact, inactive (i.e. assuming the true response rate is 0.20) and active (i.e. assuming the true response rate is 0.50) respectively. Therefore the total sample size of 25 evaluable patients will be entered. Accounting for a possible minority of patients being non-evaluable after recruitment, we aim to recruit a total of 28 patients for this study.

#### 5.5 Stratification

Response and survival analyses will be stratified between treatment naïve patients and patients who have received prior systemic treatments.



## 5.6 Concomitant Medications/Vaccinations (allowed & prohibited)

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Merck Clinical team. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician.

## 5.6.1 Acceptable Concomitant Medications

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the case report form (CRF) including all prescription, over-the-counter (OTC), herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the CRF.

All concomitant medications received within 28 days before the first dose of trial treatment and 30 days after the last dose of trial treatment should be recorded. Concomitant medications administered after 30 days after the last dose of trial treatment should be recorded for SAEs and ECIs as defined in Section 7.2.

#### 5.6.2 Prohibited Concomitant Medications

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post-complete response relapse) of this trial:

- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol
- Chemotherapy not specified in this protocol
- Investigational agents other than pembrolizumab
- Radiation therapy
  - O Note: Radiation therapy to a symptomatic solitary lesion or to the brain may be allowed at the investigator's discretion.
- Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.



• Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.

Subjects who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describes other medications, which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

#### 5.7 Rescue Medications & Supportive Care

#### **5.7.1** Supportive Care Guidelines

Subjects should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of adverse events with potential immunologic etiology are outlined below and in greater detail in the ECI guidance document. Where appropriate, these guidelines include the use of oral or intravenous treatment with corticosteroids as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the investigator determines the events to be related to pembrolizumab.

Note: if after the evaluation the event is determined not to be related, the investigator is instructed to follow the ECI reporting guidance but does not need to follow the treatment guidance (as outlined in the ECI guidance document). Refer to Section 5.2.1 for dose modification.

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event. Suggested conditional procedures, as appropriate, can be found in the ECI guidance document.

#### • Pneumonitis:

- o For **Grade 2 events**, treat with systemic corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- For Grade 3-4 events, immediately treat with intravenous steroids.
   Administer additional anti-inflammatory measures, as needed.



O Add prophylactic antibiotics for opportunistic infections in the case of prolonged steroid administration.

#### • Diarrhea/Colitis:

Subjects should be carefully monitored for signs and symptoms of enterocolitis (such as diarrhea, abdominal pain, blood or mucus in stool, with or without fever) and of bowel perforation (such as peritoneal signs and ileus).

- All subjects who experience diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion. For Grade 2 or higher diarrhea, consider GI consultation and endoscopy to confirm or rule out colitis.
- For Grade 2 diarrhea/colitis that persists greater than 3 days, administer oral corticosteroids.
- o For Grade 3 or 4 diarrhea/colitis that persists > 1 week, treat with intravenous steroids followed by high dose oral steroids.
- O When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Type 1 diabetes mellitus (if new onset, including diabetic ketoacidosis [DKA]) or ≥ Grade 3 Hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA)
  - o For **T1DM** or **Grade 3-4** Hyperglycemia
    - Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
    - Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.

### • Hypophysitis:

- For Grade 2 events, treat with corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- For **Grade 3-4** events, treat with an initial dose of IV corticosteroids followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.



### • Hyperthyroidism or Hypothyroidism:

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.

- o Grade 2 hyperthyroidism events (and Grade 2-4 hypothyroidism):
  - In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
  - In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- o Grade 3-4 hyperthyroidism
  - Treat with an initial dose of IV corticosteroid followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

#### • Hepatic:

- o For **Grade 2** events, monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with IV or oral corticosteroids
- o For **Grade 3-4** events, treat with intravenous corticosteroids for 24 to 48 hours.
- O When symptoms improve to Grade 1 or less, a steroid taper should be started and continued over no less than 4 weeks.

#### • Renal Failure or Nephritis:

- o For Grade 2 events, treat with corticosteroids.
- For Grade 3-4 events, treat with systemic corticosteroids.
- o When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

Management of Infusion Reactions: Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion.

Table 4 below shows treatment guidelines for subjects who experience an infusion reaction associated with administration of pembrolizumab (MK-3475).



Table 4 Infusion Reaction Treatment Guidelines

| NCI CTCAE Grade | Treatment | Premedication at |
|---|---|---|
| | | subsequent dosing |
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated Grade 2 Requires infusion interruption but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for < =24 hrs | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. Stop Infusion and monitor symptoms. Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDS Acetaminophen Narcotics Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. If symptoms resolve within one hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate | |
| | (e.g., from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the subject should be premedicated for the next scheduled dose. Subjects who develop Grade 2 | |
| | toxicity despite adequate premedication should be permanently discontinued from further trial treatment | |
| | administration. | |
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| | Additional appropriate medical | |
| Grade 3: | therapy may include but is not | |
| Prolonged (i.e., not | limited to: | |



| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| rapidly responsive to | IV fluids | |
| symptomatic medication | Antihistamines | |
| and/or brief interruption | NSAIDS | |
| of infusion); recurrence | Acetaminophen | |
| of symptoms following | Narcotics | |
| initial improvement; | Oxygen | |
| hospitalization indicated | Pressors | |
| for other clinical sequelae | Corticosteroids | |
| (e.g., renal impairment, | Epinephrine | |
| pulmonary infiltrates) | | |
| | Increase monitoring of vital | |
| Grade 4: | signs as medically indicated until | |
| Life-threatening; pressor | the subject is deemed medically | |
| or ventilatory support | stable in the opinion of the | |
| indicated | investigator. | |
| | Hospitalization may be | |
| | indicated. | |
| | Subject is permanently | |
| | discontinued from further trial | |
| | treatment administration. | |

Appropriate resuscitation equipment should be available in the room and a physician readily available during the period of drug administration.

### 5.8 Diet/Activity/Other Considerations

#### 5.8.1 Diet

Subjects should maintain a normal diet unless modifications are required to manage an AE such as diarrhea, nausea or vomiting.

### 5.8.2 Contraception

Pembrolizumab may have adverse effects on a fetus in utero. Furthermore, it is not known if pembrolizumab has transient adverse effects on the composition of sperm. Non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive. Highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is  $\geq$ 45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study. The two birth control methods can be



either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. Subjects should start using birth control from study Visit 1 throughout the study period up to 120 days after the last dose of study therapy.

The following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).

Subjects should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study. In order to participate in the study they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period defined in section 7.2.2-Reporting of Pregnancy and Lactation to the Sponsor and to Merck. If there is any question that a subject will not reliably comply with the requirements for contraception, that subject should not be entered into the study.

### 5.8.3 Use in Pregnancy

If a subject inadvertently becomes pregnant while on treatment with pembrolizumab, the subject will immediately be removed from the study. The site will contact the subject at least monthly and document the subject's status until the pregnancy has been completed or terminated. The outcome of the pregnancy will be reported to the Sponsor and to Merck without delay and within 24 hours to the Sponsor and within 2 working days to Merck if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn).

The study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn to the Sponsor. If a male subject impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported to the Sponsor and to Merck and followed as described above and in Section 7.2.2.

#### 5.8.4 Use in Nursing Women

It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, subjects who are breast-feeding are not eligible for enrollment.

### 5.9 Subject Withdrawal/Discontinuation Criteria

Subjects may withdraw consent at any time for any reason or be dropped from the trial at the discretion of the investigator should any untoward effect occur. In addition, a subject may be withdrawn by the investigator or the Sponsor if enrollment into the trial is inappropriate, the



trial plan is violated, or for administrative and/or other safety reasons. Specific details regarding discontinuation or withdrawal are provided in Section 7.1.4 – Other Procedures.

A subject must be discontinued from the trial for any of the following reasons:

- The subject or legal representative (such as a parent or legal guardian) withdraws consent.
- Confirmed radiographic disease progression

Note: For unconfirmed radiographic disease progression, please see Section 5.2.2

*Note*: A subject may be granted an exception to continue on treatment with confirmed radiographic progression if clinically stable or clinically improved, please see Section 7.1.2.7.1

- Unacceptable adverse experiences as described in Section 5.2.1.2
- Intercurrent illness that prevents further administration of treatment
- Investigator's decision to withdraw the subject
- The subject has a confirmed positive serum pregnancy test
- Noncompliance with trial treatment or procedure requirements
- The subject is lost to follow-up
- Completed 24 months of uninterrupted treatment with pembrolizumab or 35 administrations of study medication, whichever is later.

Note: 24 months of study medication is calculated from the date of first dose. Subjects who stop pembrolizumab after 24 months may be eligible for up to one year of additional study treatment if they progress after stopping study treatment provided they meet the requirements detailed in Section 7.1.5.5

Administrative reasons

The End of Treatment and Follow-up visit procedures are listed in Section 6 (Protocol Flow Chart) and Section 7.1.5 (Visit Requirements). After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events will be collected for 90 days after the end of treatment as described in Section 7.2.3.1). Subjects who discontinue for reasons other than progressive disease will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent or becoming lost to follow-up. After documented disease progression



each subject will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study, whichever occurs first.

## 5.9.1 Discontinuation of Study Therapy after CR

Discontinuation of treatment may be considered for subjects who have attained a confirmed CR that have been treated for at least 24 weeks with pembrolizumab and had at least two treatments with pembrolizumab beyond the date when the initial CR was declared. Subjects who then experience radiographic disease progression may be eligible for up to one year of additional treatment with pembrolizumab via the Second Course Phase at the discretion of the investigator if no cancer treatment was administered since the last dose of pembrolizumab, the subject meets the safety parameters listed in the Inclusion/Exclusion criteria, and the trial is open. Subjects will resume therapy at the same dose and schedule at the time of initial discontinuation. Additional details are provided in Section 7.1.5.5.

### 5.10 Subject Replacement Strategy

Subjects who have not received at least 2 doses of pembrolizumab shall be replaced. Final analysis of the study shall be based on intention-to-treat analysis.

## 5.11 Clinical Criteria for Early Trial Termination

Early trial termination will be the result of the criteria specified below:

- 1. Quality or quantity of data recording is inaccurate or incomplete
- 2. Poor adherence to protocol and regulatory requirements
- 3. Incidence or severity of adverse drug reaction in this or other studies indicates a potential health hazard to subjects
- 4. Plans to modify or discontinue the development of the study drug

In the event of Merck decision to no longer supply study drug, ample notification will be provided so that appropriate adjustments to subject treatment can be made.

Product: Pembrolizumab Protocol/Amendment No.:

6.0 TRIAL FLOW CHART

6.1 Study Flow Chart

| X | Screening<br>Phase | | | reatn | nent C | Treatment Cycles | | | | End of<br>Treatm<br>ent | | Post-Treatment | lent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | To | be repond 8 | To be repeated beyond 8 cycles | . 10 | | Safety | Follow I In | Survival |
| Treatment Cycle/Title: | | 1 | 2 | 'n | 4 | 5 | 9 | 7 | | Discon | dn- | Visits | Follow-Up |
| | | | | | | | | | | | | Every 6 | |
| | Main<br>Study | | | | | | | | | | | weeks post<br>discon | |
| | Screening | | | | | | | | | | | [Then | |
| | | | | | | | | | | | | every 9 | |
| | | | | | | | | | | At time | 30 days | 1 year of | |
| | | | | | - | <del></del> | | | | Jo | post | discontinua | Every 12 |
| Scheduling Window (Days): | -28 to -1 | | $\pm 3$ | ±3 | ±3 | ±3 | ±3 : | ±3 = | ±3 ] | Discon | discon | tion] | weeks |
| Administrative Procedures | | | | | | | | | | | | | 一种可能的 |
| Informed Consent | X | | | | | | | | . * | | | | |
| Inclusion/Exclusion Criteria | × | | | | | | | | | | | | |
| Demographics and Medical<br>History | × | | | | | | | | | | | | |
| Prior and Concomitant<br>Medication Review | X | X | X | × | × | × | × | × | $\times$ | × | | | |
| Trial Treatment Administration | | × | X | × | × | × | × | × | × | | | | |

Product: Pembrolizumab Protocol/Amendment No.:

Pembrolizumab in East Asian patients with acral lentiginous melanoma Version 1.2– Last updated  $9\_10\_18$ 

Product: Pembrolizumab Protocol/Amendment No.:

| X |
|---------------------|
| On-treatment Biopsy |

Product: Pembrolizumab Protocol/Amendment No.:

6.2 Second Course Phase (Retreatment with Pembrolizumab)

| | Trial Period: | | Tre | Treatment Cycles | Cycles | | | End of | | Post- | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | | | | | | | Treatment | | Treatment | |
| | Treatment Cycle: | П | 2 | m | 4 | 5 | Cycle 6 | Discon | Safety | | Survival |
| | | | | | | | and | | Follow-up | Visits | Follow-up |
| | | | | | | | peyond | | | Every 6 | |
| | | | | | | | | | | weeks | |
| | | | | | | | _ | | 30 4376 | post | |
| | | | • | | | | | At time of | oc days | discon | Every 12 |
| | | | | | | • | | discon | post<br>diccon | [Every 9 | weeks |
| | | | | | | | | | discoil | weeks | |
| | | | | | | | | | | after 1 | |
| | | - | | | • | | | | | year] | |
| Scheduli | Scheduling Window (Days) | | 1+3 | +I | +3 | +3 | ۳<br>۲+ | +3 | £ +1 | ± 7 | ± 7 |
| Administrative Procedures | अटडाब्रामस्ट | | | | | | | | | | <b>新山村</b> |
| Eligibility Criteria | | × | | | | | | | | | |
| Concomitant Medication Review | cation Review | × | × | × | × | × | × | × | × | | |
| @imical/Procedures//Assessments | ड///४ऽऽच्टऽडागाचागङ | | | | | | | | | | |
| Review Adverse Events | ents | × | × | × | × | × | × | × | × | × | |
| Full Physical Examination | nation | × | | | | | | × | | | |
| Directed Physical Examination | xamination | | × | × | × | × | × | | | | |

Pembrolizumab in East Asian patients with acral lentiginous melanoma Version 1.2- Last updated 9\_10\_18

Product: Pembrolizumab Protocol/Amendment No.:

| Vital Signs and Weight | × | × | × | × | × | × | × | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ECOG Performance Status | × | × | × | × | × | × | × | | | |
| Pembrolizumab Administration | × | × | × | × | × | × | | | | |
| Post-study Anticancer Therapy Status | | | | | | | | | × | × |
| Survival Status | | | | | | | | | | × |
| Laboratory<br>Procedures/Assessments | | | | ************************************** | | | | | | |
| Pregnancy Test [if applicable] –<br>Urine or Serum –HCG | × | | | | | | | | | |
| PT/INR and aPTT | × | | | | | | | | | |
| CBC with Differential | × | × | × | × | × | × | × | × | | |
| Chemistry Panel | × | × | × | × | × | × | × | × | | |
| Urinalysis | × | | | | | | | | | |
| T3, FT4 and TSH | × | - | × | | × | | | × | | |
| Efficacy Measurements | | | | | | | | | | |
| Tumor Imaging | × | | × | | | × | × | | × | |

**Product:** Pembrolizumab **Protocol/Amendment No.:** 

#### 7.0 TRIAL PROCEDURES

#### 7.1 Trial Procedures

The Trial Flow Chart - Section 6.0 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below. It may be necessary to perform these procedures at unscheduled time points if deemed clinically necessary by the investigator.

Furthermore, additional evaluations/testing may be deemed necessary by the Sponsor and/or Merck for reasons related to subject safety. In some cases, such evaluation/testing may be potentially sensitive in nature (e.g., HIV, Hepatitis C, etc.), and thus local regulations may require that additional informed consent be obtained from the subject. In these cases, such evaluations/testing will be performed in accordance with those regulations.

#### 7.1.1 Administrative Procedures

#### 7.1.1.1 Informed Consent

The Investigator must obtain documented consent from each potential subject prior to participating in a clinical trial.

#### 7.1.1.1.1 General Informed Consent

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

A copy of the signed and dated consent form should be given to the subject before participation in the trial.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the trial. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

Specifics about a trial and the trial population will be added to the consent form template at the protocol level.

The informed consent will adhere to IRB/ERC requirements, applicable laws and regulations and Sponsor requirements.

Product: Pembrolizumab Protocol/Amendment No.:

#### 7.1.1.2 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the trial.

### 7.1.1.3 Medical History

A medical history will be obtained by the investigator or qualified designee. Medical history will include all active conditions, and any condition diagnosed within the prior 10 years that are considered to be clinically significant by the Investigator. Details regarding the disease for which the subject has enrolled in this study will be recorded separately and not listed as medical history.

#### 7.1.1.4 Prior and Concomitant Medications Review

#### 7.1.1.4.1 Prior Medications

The investigator or qualified designee will review prior medication use, including any protocol-specified washout requirement, and record prior medication taken by the subject within 28 days before starting the trial. Treatment for the disease for which the subject has enrolled in this study will be recorded separately and not listed as a prior medication.

### 7.1.1.4.2 Concomitant Medications

The investigator or qualified designee will record medication, if any, taken by the subject during the trial. All medications related to reportable SAEs and ECIs should be recorded as defined in Section 7.2.

#### 7.1.1.5 Disease Details and Treatments

### 7.1.1.5.1 Disease Details

The investigator or qualified designee will obtain prior and current details regarding disease status.

#### 7.1.1.5.2 Prior Treatment Details

The investigator or qualified designee will review all prior cancer treatments including systemic treatments, radiation and surgeries.

### 7.1.1.5.3 Subsequent Anti-Cancer Therapy Status

The investigator or qualified designee will review all new anti-neoplastic therapy initiated after the last dose of trial treatment. If a subject initiates a new anti-cancer therapy within 30 days after the last dose of trial treatment, the 30 day Safety Follow-up visit must occur before
the first dose of the new therapy. Once new anti-cancer therapy has been initiated the subject will move into survival follow-up.

#### 7.1.2 Clinical Procedures/Assessments

# 7.1.2.1 Adverse Event (AE) Monitoring

The investigator or qualified designee will assess each subject to evaluate for potential new or worsening AEs as specified in the Trial Flow Chart and more frequently if clinically indicated. Adverse experiences will be graded and recorded throughout the study and during the follow-up period according to NCI CTCAE Version 4.0 (see Section 11.2). Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

For subjects receiving treatment with pembrolizumab all AEs of unknown etiology associated with pembrolizumab exposure should be evaluated to determine if it is possibly an event of clinical interest (ECI) of a potentially immunologic etiology (termed immunerelated adverse events, or irAEs); see the separate ECI guidance document in Appendix 4 regarding the identification, evaluation and management of potential irAEs.

Please refer to section 7.2 for detailed information regarding the assessment and recording of AEs.

## 7.1.2.2 Full Physical Exam

The investigator or qualified designee will perform a complete physical exam during the screening period. Clinically significant abnormal findings should be recorded as medical history. A full physical exam should be performed during screening,

#### 7.1.2.3 Directed Physical Exam

For cycles that do not require a full physical exam per the Trial Flow Chart, the investigator or qualified designee will perform a directed physical exam as clinically indicated prior to trial treatment administration.

### 7.1.2.4 Vital Signs

The investigator or qualified designee will take vital signs at screening, prior to the administration of each dose of trial treatment and at treatment discontinuation as specified in the Trial Flow Chart (Section 6.0). Vital signs should include temperature, pulse, respiratory rate, weight and blood pressure. Height will be measured at screening only.

#### 7.1.2.5 Eastern Cooperative Oncology Group (ECOG) Performance Scale

The investigator or qualified designee will assess ECOG status (see Section 11.1) at screening, prior to the administration of each dose of trial treatment and discontinuation of trial treatment as specified in the Trial Flow Chart.

#### 7.1.2.6 Tumor Imaging and Assessment of Disease

Tumour response will be assessed as per Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST 1.1)[11]. Treatment decisions will be based on a modification of RECIST 1.1. Specifically, patients who show evidence of disease progression (PD) at subsequent imaging, but remain clinically stable can continue on treatment at the discretion of the investigator, after which further reassessment imaging will have been done. Reassessment imaging must be done at least 4 weeks after the first assessment. If the second set of imaging shows unequivocal evidence of PD, treatment will have to be discontinued. Patients, who have discontinued treatment, either for PD or for other reasons, but have not embarked on a subsequent line of treatment, can voluntarily elect to have continual imaging at regular intervals to monitor disease status.

An exploratory correlative response assessment as per the immune-related response criteria (irRC) will also be performed.

#### 7.1.2.7 Tumor Tissue Collection and Correlative Studies Blood Sampling

Patients will require either an archival sample of their primary tumour/metastatic site for correlation studies, including PD-L1 expression as well as BRAF, c-KIT, NRAS mutational analyses. No interval systemic treatment is allowed between the time of specimen collection and start of this study. If archival samples are not available or the above tests cannot be performed on them for specific reasons, a new biopsy will have to be obtained.

Where feasible, on-treatment biopsy is also required after 2 doses of pembrolizumab for correlative studies. If the initial screening specimen was obtained from a metastatic site (either archival specimen or a dedicated screening biopsy), re-biopsy of the same site is preferable if technically feasible. Levels of PD-L1 expression in the pre- and on-treatment biopsies will be compared, and changes of which will attempt to be correlated with treatment outcomes and survival. Pathological review of the on-treatment specimen will also be performed to identify any possible changes in histopathology features (e.g. presence of lymphocyte infiltration) in the tumour during treatment, and if there are changes, whether or not this can be correlated with survival and response to treatment.

The incidence of PD-L1 expression in acral lentiginous melanoma in East Asians and its potential prognostic and predictive implications will be determined, as documented by the initial tumour specimen either from archival sample or a new biopsy. The genomic mutational landscape of acral melanomas in the East Asian population will be explored. With the mandatory on-treatment biopsy, changes in PD-L1 expression (if any) after 2 doses of

pembrolizumab can be assessed. Whether changes in PD-L1 expression in this situation may have a predictive or prognostic significance to pembrolizumab treatment will be explored.

Pharmacokinetics assessments of pembrolizumab in an East Asian population will be performed.

## 7.1.3 Laboratory Procedures/Assessments

Details regarding specific laboratory procedures/assessments to be performed in this trial are provided below. Laboratory Safety Evaluations (Hematology, Chemistry and Urinalysis)

Laboratory tests for hematology, chemistry, urinalysis, and others are specified in Table 5.

Table 5 Laboratory Tests

| Hematology | Chemistry | Urinalysis | Other |
|---|---|---|---|
| Hematocrit | Albumin | Blood | Serum β-human chorionic gonadotropin† |
| Hemoglobin | Alkaline phosphatase | Glucose | (β-hCG)† |
| Platelet count | Alanine aminotransferase (ALT) | Protein | PT (INR) |
| WBC (total and differential) Aspartate (AST) | Aspartate aminotransferase (AST) | Specific gravity | aPTT |
| Red Blood Cell Count | Lactate dehydrogenase (LDH) | Microscopic exam (If abnormal) | Total triiodothyronine (T3) |
| Absolute Neutrophil Count | Carbon Dioxide ‡ | results are noted | Free thyroxine (T4) |
| Absolute Lymphocyte Count | (CO <sub>2</sub> or biocarbonate) | Urine pregnancy test † | Thyroid stimulating hormone (TSH) |
| | Uric Acid | | PK |
| | Calcium | | |
| | Chloride | | Blood for correlative studies |
| | Glucose | | |
| | Phosphorus | | |
| | Potassium | | |
| | Sodium | | |
| | Magnesium | | |
| | Total Bilirubin | | |
| | Direct Bilirubin (If total bilirubin is elevated above the upper limit of normal) | | |

Pembrolizumab in East Asian patients with acral lentiginous melanoma Version 1.2– Last updated 9\_10\_18

Product: Pembrolizumab Protocol/Amendment No.:

| ſ | | | | |
|---|---|---|---|---|
| | er | | | srum pregnancy |
| | Other | | | ed as negative, a se |
| | Urinalysis | | | otential only. If urine pregnancy results cannot be confirmed as negative, a serum pregnancy |
| | Chemistry | Total protein | Blood Urea Nitrogen | nildbearing potential only. If urine pre |
| | Hematology | | | † Perform on women of childbearing po |

‡ If considered standard of care in your region.

test will be required.

Pembrolizumab in East Asian patients with a cral lentiginous melanoma Version 1.2– Last updated  $9\_10\_18$ 

Laboratory tests for screening or entry into the Second Course Phase should be performed within 10 days prior to the first dose of treatment. After Cycle 1, pre-dose laboratory procedures can be conducted up to 72 hours prior to dosing. Results must be reviewed by the investigator or qualified designee and found to be acceptable prior to each dose of trial treatment.

#### 7.1.3.1 Pharmacokinetic/Pharmacodynamic Evaluations

#### 7.1.3.1.1 Blood Collection for Serum Pembrolizumab

Sample collection, storage and shipment instructions for serum samples will be provided in the Laboratory Manual.

The time-points for PK blood sampling are described in Section 6 – Trial Flow Chart.

#### 7.1.3.1.2 Blood Collection for Anti-Pembrolizumab Antibodies

Sample collection, storage and shipment instructions for blood samples will be provided in the Laboratory Manual.

#### 7.1.3.2 Correlative studies

#### 7.1.3.2.1 PD-L1 expression in archival sample and on-treatment biopsy

PD-L1 expression testing will be performed in a centralized facility (QualTek). Shipping and preparatory details can be found in the laboratory manual.

- Formalin fixed paraffin embedded tissue samples are acceptable; a fine needle aspirate, frozen sample, plastic embedded sample, cell block, clot, bone, bone marrow or cytologic specimen will not be acceptable for IHC analysis.
- It is recommended that FFPE blocks be sectioned fresh (within 7 days of sectioning and sending for PD-L1 analysis) onto positively charged slides; slides should be stored and shipped at 2-8C in the dark.
- Recommended fixation time for samples is 24 hours to 48 hours in 10% neutral buffered formalin.

#### 7.1.3.2.2. Mutational analysis of BRAF, NRAS and KIT

Mutations on BRAF exon 11 and 15, NRAS exons 1 and 2, and KIT exons 9,11,13,17 and 18 are screened by PCR-direct sequencing.

Tumor cells are isolated from paraffin sections by manual microdissection. Genomic DNA is extracted for the PCR amplification. The PCR products are purified with 1  $\mu$ l ExoI/SAP (37°C for 15 minutes, then 85°C for 15 minutes) and then sequenced directly on both strands

using the BigDye® Terminator v1.1 cycle sequencing kit (Applied Biosystems) according to manufacturer's protocol and analyzed by the Life Technologies 3500 Genetic Analyzer. Positive and negative controls are included. The data are collected and analyzed using Applied Biosystem sequencing analysis software. All mutations are re-confirmed by independent PCR reactions and direct sequencing.

#### 7.1.4 Other Procedures

#### 7.1.4.1 Withdrawal/Discontinuation

When a subject discontinues/withdraws prior to trial completion, all applicable activities scheduled for the final trial visit should be performed at the time of discontinuation. Any adverse events which are present at the time of discontinuation/withdrawal should be followed in accordance with the safety requirements outlined in Section 7.2 - Assessing and Recording Adverse Events. Subjects who a) attain a CR or b) complete 24 months of treatment with pembrolizumab may discontinue treatment with the option of restarting treatment if they meet the criteria specified in Section 7.1.5.5. After discontinuing treatment following assessment of CR, these subjects should return to the site for a Safety Follow-up Visit (described in Section 7.1.5.3.1) and then proceed to the Follow-Up Period of the study (described in Section 7.1.5.4).

# 7.1.5 Visit Requirements

Visit requirements are outlined in Section 6.0 - Trial Flow Chart. Specific procedure-related details are provided above in Section 7.1 - Trial Procedures.

#### 7.1.5.1 Screening

#### 7.1.5.1.1 Screening Period

The screening period will be a duration of 28 days thereafter, inclusive of the date of consenting.

#### 7.1.5.2 Treatment Period

Approximately 28 patients biologics-naïve accrual lentiginous melanoma patients shall be enrolled to evaluate the anti-tumor activity and further assess the safety, tolerability of pembrolizumab in this population.

#### 7.1.5.3 Post-Treatment Visits

#### 7.1.5.3.1 Safety Follow-Up Visit

The mandatory Safety Follow-Up Visit should be conducted approximately 30 days after the last dose of trial treatment or before the initiation of a new anti-cancer treatment, whichever comes first. All AEs that occur prior to the Safety Follow-Up Visit should be recorded.

Subjects with an AE of Grade > 1 will be followed until the resolution of the AE to Grade 0-1 or until the beginning of a new anti-neoplastic therapy, whichever occurs first. SAEs that occur within 90 days of the end of treatment or before initiation of a new anti-cancer treatment should also be followed and recorded. Subjects who are eligible for retreatment with pembrolizumab (as described in Section 7.1.5.5) may have up to two safety follow-up visits, one after the Treatment Period and one after the Second Course Phase.

#### 7.1.5.4 Follow-up Visits

Subjects who discontinue trial treatment for a reason other than disease progression will move into the Follow-Up Phase and should be assessed every 6 weeks ( $42 \pm 7$  days) by radiologic imaging to monitor disease status. After 1 year, the imaging time point will occur every 9 weeks ( $\pm$  7 days). Every effort should be made to collect information regarding disease status until the start of new anti-neoplastic therapy, disease progression, death, end of the study or if the subject begins retreatment with pembrolizumab as detailed in Section 7.1.5.5. Information regarding post-study anti-neoplastic treatment will be collected if new treatment is initiated.

Subjects who are eligible to receive retreatment with pembrolizumab according to the criteria in Section 7.1.5.5 will move from the follow-up phase to the Second Course Phase when they experience disease progression. Details are provided in Section 6.2 – Trial Flow Chart for Retreatment.

#### 7.1.5.4.1 Survival Follow-up

Once a subject experiences confirmed disease progression or starts a new anti-cancer therapy, the subject moves into the survival follow-up phase and should be contacted by telephone every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.

#### 7.1.5.5 Second Course Phase (Retreatment Period)

Subjects who stop pembrolizumab with SD or better may be eligible for up to one year of additional pembrolizumab therapy if they progress after stopping study treatment. This retreatment is termed the Second Course Phase of this study and is only available if the study remains open and the subject meets the following conditions:

#### Either

- Stopped initial treatment with pembrolizumab after attaining an investigatordetermined confirmed CR according to RECIST 1.1, and
  - Was treated for at least 24 weeks with pembrolizumab before discontinuing therapy

 Received at least two treatments with pembrolizumab beyond the date when the initial CR was declared

#### OR

 Had SD, PR or CR and stopped pembrolizumab treatment after 24 months of study therapy for reasons other than disease progression or intolerability

#### AND

- Experienced an investigator-determined confirmed radiographic disease progression after stopping their initial treatment with pembrolizumab
- Did not receive any anti-cancer treatment since the last dose of pembrolizumab
- Has a performance status of 0 or 1 on the ECOG Performance Scale
- Demonstrates adequate organ function as detailed in Section 5.1.2
- Female subject of childbearing potential should have a negative serum or urine pregnancy test within 72 hours prior to receiving retreatment with study medication.
- Female subject of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of child bearing potential are those who have not been surgically sterilized or have been free from menses for > 1 year.
- Male subject should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
- Does not have a history or current evidence of any condition, therapy, or laboratory abnormality that might interfere with the subject's participation for the full duration of the trial or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Subjects who restart treatment will be retreated at the same dose and dose interval as when they last received pembrolizumab. Treatment will be administered for up to one additional year.

Visit requirements are outlined in Section 6.0 - Trial Flow Chart.

#### 7.2 Assessing and Recording Adverse Events

An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Merck's product, is also an adverse event.

Changes resulting from normal growth and development that do not vary significantly in frequency or severity from expected levels are not to be considered adverse events. Examples of this may include, but are not limited to, teething, typical crying in infants and children and onset of menses or menopause occurring at a physiologically appropriate time.

Merck product includes any pharmaceutical product, biological product, device, diagnostic agent or protocol-specified procedure, whether investigational (including placebo or active comparator medication) or marketed, manufactured by, licensed by, provided by or distributed by Merck for human use.

Adverse events may occur during the course of the use of Merck product in clinical trials or within the follow-up period specified by the protocol, or prescribed in clinical practice, from overdose (whether accidental or intentional), from abuse and from withdrawal.

Adverse events may also occur in screened subjects during any pre-allocation baseline period as a result of a protocol-specified intervention, including washout or discontinuation of usual therapy, diet, placebo treatment or a procedure.

Progression of the cancer under study is not considered an adverse event unless it is considered to be drug related by the investigator.

All adverse events will be recorded from the time the consent form is signed through 30 days following cessation of treatment and at each examination on the Adverse Event case report forms/worksheets. The reporting timeframe for adverse events meeting any serious criteria is described in section 7.2.3.1.

# 7.2.1 Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor and to Merck

For purposes of this trial, an overdose of pembrolizumab will be defined as any dose of 1,000 mg or greater (≥5 times the indicated dose). No specific information is available on the treatment of overdose of pembrolizumab. Appropriate supportive treatment should be provided if clinically indicated. In the event of overdose, the subject should be observed

closely for signs of toxicity. Appropriate supportive treatment should be provided if clinically indicated.

If an adverse event(s) is associated with ("results from") the overdose of a Merck product, the adverse event(s) is reported as a serious adverse event, even if no other seriousness criteria are met.

If a dose of Merck's product meeting the protocol definition of overdose is taken without any associated clinical symptoms or abnormal laboratory results, the overdose is reported as a non-serious Event of Clinical Interest (ECI), using the terminology "accidental or intentional overdose without adverse effect."

All reports of overdose with and without an adverse event must be reported within 24 hours to the Sponsor and within 2 working days hours to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

#### 7.2.2 Reporting of Pregnancy and Lactation to the Sponsor and to Merck

Although pregnancy and lactation are not considered adverse events, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject (spontaneously reported to them), including the pregnancy of a male subject's female partner that occurs during the trial or within 120 days of completing the trial completing the trial, or 30 days following cessation of treatment if the subject initiates new anticancer therapy, whichever is earlier. All subjects and female partners of male subjects who become pregnant must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, benign hydatidiform mole, blighted ovum, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events (Important Medical Events). If the pregnancy continues to term, the outcome (health of infant) must also be reported.

Such events must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)

## 7.2.3 Immediate Reporting of Adverse Events to the Sponsor and to Merck

#### 7.2.3.1 Serious Adverse Events

A serious adverse event is any adverse event occurring at any dose or during any use of Merck's product that:

- Results in death;
- Is life threatening;
- Results in persistent or significant disability/incapacity;
- Results in or prolongs an existing inpatient hospitalization;
- Is a congenital anomaly/birth defect;

- Is a new cancer (that is not a condition of the study);
- Is associated with an overdose;
- Is an other important medical event

Refer to Table 6 for additional details regarding each of the above criteria.

Any serious adverse event, or follow up to a serious adverse event, including death due to any cause other than progression of the cancer under study that occurs to any subject from the time the consent is signed through 90 days following cessation of treatment, or the initiation of new anti-cancer therapy, whichever is earlier, whether or not related to Merck product, must be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety.

Non-serious Events of Clinical Interest will be forwarded to Merck Global Safety and will be handled in the same manner as SAEs.

Additionally, any serious adverse event, considered by an investigator who is a qualified physician to be related to Merck product that is brought to the attention of the investigator at any time outside of the time period specified in the previous paragraph also must be reported immediately to the Sponsor and to Merck.

# SAE reports and any other relevant safety information are to be forwarded to the Merck Global Safety facsimile number: +1-215-993-1220

A copy of all 15 Day Reports and Annual Progress Reports is submitted as required by FDA, European Union (EU), Pharmaceutical and Medical Devices agency (PMDA) or other local regulators. Investigators will cross reference this submission according to local regulations to the Merck Investigational Compound Number (IND, CSA, etc.) at the time of submission. Additionally investigators will submit a copy of these reports to Merck & Co., Inc. (Attn: Worldwide Product Safety; FAX 215 993-1220) at the time of submission to FDA.

All subjects with serious adverse events must be followed up for outcome.

#### 7.2.3.2 Events of Clinical Interest

Selected non-serious and serious adverse events are also known as Events of Clinical Interest (ECI) and must be recorded as such on the Adverse Event case report forms/worksheets and reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220)Events of clinical interest for this trial include:

1. an overdose of Merck product, as defined in Section 7.2.1 - Definition of an Overdose for This Protocol and Reporting of Overdose to the Sponsor, that is not associated with clinical symptoms or abnormal laboratory results.

2. an elevated AST or ALT lab value that is greater than or equal to 3X the upper limit of normal and an elevated total bilirubin lab value that is greater than or equal to 2X the upper limit of normal and, at the same time, an alkaline phosphatase lab value that is less than 2X the upper limit of normal, as determined by way of protocol-specified laboratory testing or unscheduled laboratory testing.\*

\*Note: These criteria are based upon available regulatory guidance documents. The purpose of the criteria is to specify a threshold of abnormal hepatic tests that may require an additional evaluation for an underlying etiology. The trial site guidance for assessment and follow up of these criteria can be found in the Investigator Trial File Binder (or equivalent).

#### 1. Additional adverse events:

A separate guidance document has been provided entitled "Event of Clinical Interest Guidance Document" (previously entitled, "Event of Clinical Interest and Immune-Related Adverse Event Guidance Document"). This document can be found in Appendix 4 and provides guidance regarding identification, evaluation and management of ECIs and irAEs.

ECIs (both non-serious and serious adverse events) identified in this guidance document from the date of first dose through 90 days following cessation of treatment, or 30 days after the initiation of a new anticancer therapy, whichever is earlier, need to be reported within 24 hours to the Sponsor and within 2 working days to Merck Global Safety. (Attn: Worldwide Product Safety; FAX 215 993-1220), regardless of attribution to study treatment, consistent with standard SAE reporting guidelines.

Subjects should be assessed for possible ECIs prior to each dose. Lab results should be evaluated and subjects should be asked for signs and symptoms suggestive of an immune-related event. Subjects who develop an ECI thought to be immune-related should have additional testing to rule out other etiologic causes. If lab results or symptoms indicate a possible immune-related ECI, then additional testing should be performed to rule out other etiologic causes. If no other cause is found, then it is assumed to be immune-related.

#### 7.2.4 Evaluating Adverse Events

An investigator who is a qualified physician will evaluate all adverse events according to the NCI Common Terminology for Adverse Events (CTCAE), version 4.0. Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

All adverse events regardless of CTCAE grade must also be evaluated for seriousness.

Table 6 Evaluating Adverse Events

An investigator who is a qualified physician, will evaluate all adverse events as to:

| V4.0 | Grade 1 | Mild; asymptomatic or mid symptoms; clinical or diagnostic observations only; intervention |
|---|---|---|
| CTCAE<br>Grading | | not indicated. |
| | Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. |
| | Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation or hospitalization indicated; disabling; limiting self-care ADL. |
| | Grade 4 | Life threatening consequences; urgent intervention indicated. |
| | Grade 5 | Death related to AE |
| Seriousness | A serious adv | A serious adverse event is any adverse event occurring at any dose or during any use of Merck product that: |
| | +Results in death; or | eath; or |
| | †Is life threatening; or | tening; or places the subject, in the view of the investigator, at immediate risk of death from the event |
| | as it occurred (Note: Th | (Note: This does not include an adverse event that, had it occurred in a more severe form, might have |
| | caused death.); or | ); or |
| | †Results in a | *Results in a persistent or significant disability/incapacity (substantial disruption of one's ability to conduct |
| | normal life functions); or | nctions); or |
| | +Results in o | *Results in or prolongs an existing inpatient hospitalization (hospitalization is defined as an inpatient |
| | admission, re | admission, regardless of length of stay, even if the hospitalization is a precautionary measure for continued |
| | observation. ( | observation. (Note: Hospitalization [including hospitalization for an elective procedure] for a preexisting condition |
| | which has not worsened | t worsened does not constitute a serious adverse event.); or |
| | †Is a congeni | †Is a congenital anomaly/birth defect (in offspring of subject taking the product regardless of time to |
| | diagnosis);or | |
| | Is a new can | Is a new cancer; (that is not a condition of the study) or |
| | Is an overdo | Is an overdose (whether accidental or intentional). Any adverse event associated with an overdose is considered a |
| | serious adver | serious adverse event. An overdose that is not associated with an adverse event is considered a non-serious event of |
| | clinical intere | clinical interest and must be reported within 24 hours. |

| | Other impormay be considerable | Other important medical events that may not result in death, not be life threatening, or not require hospitalization may be considered a serious adverse event when, based upon appropriate medical judgment, the event may |
|---|---|---|
| | jeopardize the previously (de | jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed previously (designated above by a †). |
| Duration | Record the staunits | Record the start and stop dates of the adverse event. If less than 1 day, indicate the appropriate length of time and units |
| Action | Did the adver | Did the adverse event cause the Merck product to be discontinued? |
| taken | | |
| Relationship | Did the Merck product | k product cause the adverse event? The determination of the likelihood that the Merck product caused |
| to test drug | the adverse event will | vent will be provided by an investigator who is a qualified physician. The investigator's signed/dated |
| | initials on the | initials on the source document or worksheet that supports the causality noted on the AE form, ensures that a |
| | medically qua | medically qualified assessment of causality was done. This initialed document must be retained for the required |
| | regulatory tin | regulatory time frame. The criteria below are intended as reference guidelines to assist the investigator in assessing |
| | the likelihood | the likelihood of a relationship between the test drug and the adverse event based upon the available information. |
| | The followin | The following components are to be used to assess the relationship between the Merck product and the AE; |
| | the greater the | the greater the correlation with the components and their respective elements (in number and/or intensity), the more |
| | likely the Me | likely the Merck product caused the adverse event (AE): |
| | Exposure | Is there evidence that the subject was actually exposed to the Merck product such as: reliable history, |
| | ı | acceptable compliance assessment (pill count, diary, etc.), expected pharmacologic effect, or |
| | | measurement of drug/metabolite in bodily specimen? |
| | Time | Did the AE follow in a reasonable temporal sequence from administration of the Merck product? |
| | Course | Is the time of onset of the AE compatible with a drug-induced effect (applies to trials with |
| | | investigational medicinal product)? |
| | Likely | Is the AE not reasonably explained by another etiology such as underlying disease, other |
| | Cause | drug(s)/vaccine(s), or other host or environmental factors |

| Relationship | The following compo | g components are to be used to assess the relationship between the test drug and the AE: |
|---|---|---|
| to Merck | Dechallenge | Was the Merck product discontinued or dose/exposure/frequency reduced? |
| product | | If yes, did the AE resolve or improve? |
| (continued) | | If yes, this is a positive dechallenge. If no, this is a negative dechallenge. |
| | | (Note: This criterion is not applicable if: (1) the AE resulted in death or permanent disability; (2) the |
| | | AE resolved/improved despite continuation of the Merck product; or (3) the trial is a single-dose |
| | | drug trial); or (4) Merck product(s) is/are only used one time.) |
| | Rechallenge | Was the subject re-exposed to the Merck product in this study? |
| | | If yes, did the AE recur or worsen? |
| | | If yes, this is a positive rechallenge. If no, this is a negative rechallenge. |
| | | (Note: This criterion is not applicable if: (1) the initial AE resulted in death or permanent disability, |
| | | or (2) the trial is a single-dose drug trial); or (3) Merck product(s) is/are used only one time). |
| | | NOTE: IF A RECHALLENGE IS PLANNED FOR AN ADVERSE EVENT WHICH WAS |
| | | SERIOUS AND WHICH MAY HAVE BEEN CAUSED BY THE MERCK PRODUCT, OR IF |
| | | REEXPOSURE TO THE MERCK PRODUCT POSES ADDITIONAL POTENTIAL |
| | | SIGNIFICANT RISK TO THE SUBJECT, THEN THE RECHALLENGE MUST BE APPROVED |
| | | IN ADVANCE BY THE U.S. CLINICAL MONITOR AS PER DOSE MODIFICATION |
| | | GUIDELINES IN THE PROTOCOL. |
| | Consistency | Is the clinical/pathological presentation of the AE consistent with previous knowledge regarding the |
| | with Trial | Merck product or drug class pharmacology or toxicology? |
| | Treatment | |
| | Profile | |
| The assessmer | The assessment of relationship will be | be will be reported on the case report forms /worksheets by an investigator who is a qualified physician |
| according to h | is/her best clini | according to his/her best clinical judgment, including consideration of the above elements. |
| Record one of the | f the | Use the following scale of criteria as guidance (not all criteria must be present to be indicative |
| following | | of a Merck product relationship). |

Product: MK-3475 Protocol/Amendment No.:

| Yes, there is a reasonable | ble There is evidence of exposure to the Merck product. The temporal sequence of the AE onset relative |
|---|---|
| possibility of Merck | to the administration of the Merck product is reasonable. The AE is more likely explained by the |
| product relationship. | Merck product than by another cause. |
| No, there is not a | Subject did not receive the Merck product OR temporal sequence of the AE onset relative to |
| reasonable possibility | administration of the Merck product is not reasonable OR there is another obvious cause of the AE. |
| Merck product | (Also entered for a subject with overdose without an associated AE.) |
| relationship | |

Table 8 Dose Modification and Toxicity Management Guidelines for Immune-related AEs Associated with Pembrolizumab

| | V. Do Sell Sell-Mediane | | | · | |
|---|---|---|---|---|---|
| itiated upon AE improving to Grade 1 or less and continue to taper over at least 4 weeks. mab has been withheld, pembrolizumab can be resumed after AE has been reduced to Grade 1 or 0 and Pembrolizumab should be permanently discontinued if AE does not resolve within 12 weeks of last dose or ito <10 mg prednisone or equivalent per day within 12 weeks. AEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosuppressive treatment of be controlled by corticosteroids. | Monitor and follow-up | <ul> <li>Monitor participants for signs and symptoms of pneumonitis</li> <li>Evaluate participants with suspected</li> </ul> | pneumonnus with rathographic infaging and initiate corticosteroid treatment Add prophylactic antibiotics for opportunistic infections | <ul> <li>Monitor participants for signs and symptoms of enterocolitis (ie, diarrhea, abdominal pain, blood or mucus in stool with or without fever) and of bowel perforation (ie, peritoneal signs and ileus).</li> <li>Participants with &gt; Grade 2 diarrhea</li> </ul> | <ul> <li>suspecting contasts should consider Officers consultation and performing endoscopy to rule out colitis.</li> <li>Participants with diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be</li> </ul> |
| trated upon AE improving to Grade I or less and continue to taper over at least 4 weeks has been withheld, pembrolizumab can be resumed after AE has been reduced to Greenbrolizumab should be permanently discontinued if AE does not resolve within 12 we to ≤10 mg prednisone or equivalent per day within 12 weeks. AEs, IV corticosteroid should be initiated first followed by oral steroid. Other immunosit be controlled by corticosteroids. | irAE management with<br>corticosteroid and/or other<br>therapies | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | | Administer corticosteroids (initial<br>dose of 1-2 mg/kg prednisone or<br>equivalent) followed by taper | |
| instructions: Corticosteroid taper should be initiated upon AE improving to Grad For situations where pembrolizumab has been withheld, pembrolizucorticosteroid has been tapered. Pembrolizumab should be permane corticosteroids caunot be reduced to ≤10 mg prednisone or equivale. For severe and life-threatening irAEs, IV corticosteroid should be in should be initiated if itAEs cannot be controlled by corticosteroids. | Action taken to<br>pembrolizumab | Withhold | Permanently<br>discontinue | Withhold | Permanently<br>discontinue |
| instructions: Corticosteroid taper should be ini For situations where pembrolizur corticosteroid has been tapered. F corticosteroids camot be reduced For severe and life-threatening ir, should be initiated if it AEs canno | Toxicity grade or conditions (CTCAEv4:0) | Grade 2 | Grade 3 or 4, or recurrent Grade 2 | Grade 2 or 3 | Grade 4 |
| General instructions: 1. Corticosteroid 2. For situations corticosteroid l corticosteroids 3. For severe and should be initia | Immune-related<br>AEs | Pneumonitis | | Diarrhea / Colitis | |

Pembrolizumab in East Asian patients with a cral lentiginous melanoma Version 1.2– Last updated 9\_10\_18

Product: MK-3475 Protocol/Amendment No.:

| | | | | | | | | | | —————————————————————————————————————— | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| substituted via IV infusion. | Monitor with liver function tests (consider weekly or more frequently until liver enzyme value returned to baseline or is | stable | Monitor participants for hyperglycemia or other signs and symptoms of diabetes. | | | Monitor for signs and symptoms of hypophysitis (including hypopituitarism and adrenal insufficiency) | | Monitor for signs and symptoms of thyroid disorders. | | Monitor for signs and symptoms of thyroid disorders. | Monitor changes of renal function |
| <u> </u> | • | S | • | | | • | | • | | • | • |
| | Administer corticosteroids (initial dose of 0.5- 1 mg/kg prednisone or equivalent) followed by taper | Administer corticosteroids (initial dose of 1-2 mg/kg prednisone or equivalent) followed by taper | Initiate insulin replacement therapy for participants with | Administer anti-hyperglycemic in participants with hyperglycemia | | <ul> <li>Administer corticosteroids and<br/>initiate hormonal replacements as<br/>clinically indicated.</li> </ul> | | • Treat with non-selective beta-<br>blockers (eg, propranolol) or<br>thionamides as appropriate | | Initiate thyroid replacement hormones (eg, levothyroxine or liothyroinine) per standard of care | Administer corticosteroids |
| | Withhold | Permanently<br>discontinue | Withhold | | | Withhold | Withhold or permanently discontinue | Continue | Withhold or permanently discontinue | Continue | Withhold |
| | Grade 2 | Grade 3 or 4 | Newly onset<br>TIDM or | Orade 5 or 4 hyperglycemia associated with evidence of β-cell | failure | Grade 2 | Grade 3 or 4 | Grade 2 | Grade 3 or 4 | Grade 2-4 | Grade 2 |
| | AST / ALT<br>elevation or<br>Increased | bilirubin | Type 1 diabetes mellitus (T1DM) | or<br>Hyperglycemia | | Hypophysitis | | Hyperthyroidism | | Hypothyroidism | Nephritis and<br>Renal |

Product: MK-3475
Protocol/Amendment No.:

For participants with Grade 3 or 4 immune-related endocrinopathy where withhold of pembrolizumab is required, pembrolizumab may be resumed when AE resolves to  $\leq$  Grade 2 and is controlled with hormonal replacement therapy or achieved metabolic control (in case of T1DM). 1. Withhold or permanently discontinue pembrolizumab is at the discretion of the investigator or treating physician. NOTE:

**Product:** MK-3475

Protocol/Amendment No.:

# 7.2.5 Sponsor Responsibility for Reporting Adverse Events

All Adverse Events will be reported to regulatory authorities, IRB/IECs and investigators in accordance with all applicable global laws and regulations.

#### 8.0 STATISTICAL ANALYSIS PLAN

#### 8.1 Statistical Analysis Plan Summary

#### **8.1.1** Definition of Endpoints

The study population for all analyses (intent-to-treat population), except for the analysis of ORR, DR, CBR, TTP, and PFS, will be defined as all patients enrolled in the study that receive at least 1 dose of study medication. The set of patients to be analyzed for ORR, DR, CBR, TTP, and PFS, is all patients with measurable disease at baseline, receiving at least one dose of pembrolizumab with a response assessment made by the Investigator (evaluable population). The analysis of the primary endpoint will consider patients who do not have onstudy radiographic tumor re-evaluation as non-responders in the assessment of objective tumor response rate. Endpoints calculated and their definitions include the following:

- ORR is defined as the proportion of patients with confirmed complete response (CR) or confirmed partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST), relative to the total evaluable patient population.
- CBR is defined as the percent of patients with confirmed CR, PR, or stable disease for >/= 6 months on study according to RECIST 1.1, relative to the total evaluable patient population.
- TTP defined as the time from start of study (Cycle 1) to first documentation of objective tumor progression. TTP data will be censored on the day following the date of the last tumor assessment documenting absence of progressive disease for patients who do not have objective tumor progression and are still on study at the time of an analysis, are given antitumor treatment other than the study treatment, are removed from study follow-up prior to documentation of objective tumor progression. Patients lacking an evaluation of tumor response after their first dose will have their event time censored at Day 1.
- PFS is defined as the time from start of study treatment to first documentation of objective tumor progression, or to death due to any cause. PFS data will be censored on the day following the date of the last tumor assessment documenting absence of progressive disease for patients who do not have objective tumor progression and are still on study at the time of an analysis, are given anti-tumor treatment other than the study treatment, or are removed from study follow-up prior to documentation of objective tumor progression. Patients lacking an evaluation of tumor response after their first dose will have their event time censored at Day 1.

• OS is defined as the time from start of study treatment to date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the patient is known to be alive. Patients lacking data beyond the day of first dose will have their survival times censored at 1 day.

Descriptive statistics will be used to summarize all patient characteristics, diagnoses, treatment administration/compliance, activity endpoints, safety parameters, and cancer biomarkers. The ORR will be provided along with the corresponding exact 95% 2-sided confidence interval using standard methods based on the binomial distribution. Time-to-event data will be summarized using the method of Kaplan-Meier. Data will also be displayed graphically, where appropriate.

#### 8.1.2 Rationale for current sample size calculation

The primary objective is to determine the ORR (CR+PR) of pembrolizumab in patients with acral lentiginous melanoma who have not received PD-1/PD-L1 inhibitors. Based on literature review, the ORR of first line treatment with checkpoint inhibitors of melanoma in general is in the range of 32-40%.

We assume that the ORR achievable with pembrolizumab in acral lentiginous melanoma would be similar.

The Simon's Minimax two-stage phase II design was used to calculate sample size. We consider the pembrolizumab to be inactive if the treatment response rate (confirmed CR and PR) is  $\leq 10\%$ , and consider the pembrolizumab as active if the treatment response rate is  $\geq 30\%$ . Therefore, assuming  $P_0 = 0.10$ ,  $P_1 = 0.30$ , and the type I error of 0.05 with power of 80%, the sample size and stopping rule are as follow:

Stage I: Accrue 15 patients; if 1 or less of the 15 patients are non-responders, we would stop the study and conclude pembrolizumab as inactive, otherwise proceed to stage II.

Stage II: Accrue an additional 10 patients. If 5 or less of the 25 patients are non-responders, pembrolizumab will be deemed inactive.

Using this phase II design the average sample size is 19.5 patients if the treatment is in fact, inactive (i.e. assuming the true response rate is 0.20) and active (i.e. assuming the true response rate is 0.50) respectively. Therefore the total sample size of 25 evaluable patients will be entered. Accounting for a possible minority of patients being non-evaluable after recruitment, we aim to recruit a total of 28 patients for this study.

#### 8.1.3 Interim Analysis

After accrual of the first 15 patients, an interim analysis will be performed for futility assessment before proceeding to stage II.

#### 8.2 Population for Analyses

- All enrolled subjects: All subjects who sign an informed consent form
- All treated subjects: All subjects who receive at least one dose of study medication
- Pharmacokinetic subjects: All subjects who receive at least one dose of study of medication and have available serum concentration data
- Response evaluable subjects: All subjects who receive at least one dose of study medication, and i) have measureable disease at baseline, and ii) have at least one screening (i.e. baseline) and one on-study tumor assessment or documented clinical disease progression/death.

# 9.0 LABELING, PACKAGING, STORAGE AND RETURN OF CLINICAL SUPPLIES

## 9.1 Investigational Product

The investigator shall take responsibility for and shall take all steps to maintain appropriate records and ensure appropriate supply, storage, handling, distribution and usage of investigational product in accordance with the protocol and any applicable laws and regulations.

Clinical Supplies will be provided by Merck as summarized in Table 7.

Table 7 Product Descriptions

| Product Name & Potency | Dosage Form |
|---------------------------|------------------------|
| Pembrolizumab 100 mg/ 4mL | Solution for Injection |

Product: MK-3475

Protocol/Amendment No.:

#### 9.2 Packaging and Labeling Information

Clinical supplies will be affixed with a clinical label in accordance with regulatory requirements.

#### 9.3 Clinical Supplies Disclosure

This trial is open-label; therefore, the subject, the trial site personnel, the Sponsor and/or designee are not blinded to treatment. Drug identity (name, strength) is included in the label text; random code/disclosure envelopes or lists are not provided.

#### 9.4 Storage and Handling Requirements

Clinical supplies must be stored in a secure, limited-access location under the storage conditions specified on the label.

Receipt and dispensing of trial medication must be recorded by an authorized person at the trial site.

Clinical supplies may not be used for any purpose other than that stated in the protocol.

#### 9.5 Returns and Reconciliation

The investigator is responsible for keeping accurate records of the clinical supplies received from Merck or designee, the amount dispensed to and returned by the subjects and the amount remaining at the conclusion of the trial.

Upon completion or termination of the study, all unused and/or partially used investigational product will be destroyed at the site per institutional policy. It is the Investigator's responsibility to arrange for disposal of all empty containers, provided that procedures for proper disposal have been established according to applicable federal, state, local and institutional guidelines and procedures, and provided that appropriate records of disposal are kept.

#### 10.0 ADMINISTRATIVE AND REGULATORY DETAILS

#### 10.1 Ethical considerations and administrative procedures

This clinical study was designed, shall be implemented and reported in accordance with the ICH Harmonized Tripartite Guidelines for Good Clinical Practice, with applicable local regulations (including European Directive 2001/20/EC and US Code of Federal Regulations Title 21), and with the ethical principles laid down in the Declaration of Helsinki.

**Product:** MK-3475

Protocol/Amendment No.:

# 10.2 Responsibilities of the investigator and IRB/IEC/REB

The protocol and the proposed informed consent form must be reviewed and approved by a properly constituted Institutional Review Board/Independent Ethics Committee/Research Ethics Board (IRB/IEC/REB) before study start. Prior to study start, the investigator is required to sign a protocol signature page confirming his/her agreement to conduct the study in accordance with these documents and all of the instructions and procedures found in this protocol.

# 10.3 Study documentation, record keeping and retention of records

Participating site(s) will maintain appropriate medical and research records for this trial, in compliance with Section 4.9 of the ICH E6 GCP, and regulatory and institutional requirements for the protection of confidentiality of patients.

Source data are all information, original records of clinical findings, observations, or other activities in a clinical trial necessary for the reconstruction and evaluation of the trial. Examples of these original documents and data records include, but are not limited to, hospital records, clinical and office charts, laboratory notes, memoranda, patients' diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, photographic negatives, microfilm or magnetic media, x-rays, and patient files and records kept at the pharmacy, at the laboratories, and medico-technical departments involved in the clinical trial.

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site Principal Investigator. The study case report form (CRF) is the primary data collection instrument for the study. The investigator should ensure the accuracy, completeness, legibility, and timeliness of the data reported in the CRFs and all other required reports. Data reported on the CRF, that are derived from source documents, should be consistent with the source documents or the discrepancies should be explained. All data requested on the CRF must be recorded. Any missing data must be explained. Any change or correction to a paper CRF should be dated, initialed, and explained (if necessary) and should not obscure the original entry. For electronic CRFs an audit trail will be maintained by the system.

The investigator should retain records of the changes and corrections to paper CRFs. The investigator/institution should maintain the trial documents as specified in Essential Documents for the Conduct of a Clinical Trial (ICH E6 Section 8) and as required by applicable regulations and/or guidelines. The investigator/institution should take measures to prevent accidental or premature destruction of these documents.

Essential documents (written and electronic) should be retained for a period of not less than fifteen (15) years from the completion of the Clinical Trial unless Sponsor provides written permission to dispose of them or, requires their retention for an additional period of time because of applicable laws, regulations and/or guidelines.

#### 10.4 Confidentiality

The investigator must ensure anonymity of the patients; patients must not be identified by names in any documents submitted. Signed informed consent forms and patient enrollment log must be kept strictly confidential to enable patient identification at the site.

#### 10.5 Compliance with Financial Disclosure Requirements

Financial disclosures should be provided by study personnel who are directly involved in the treatment or evaluation of patients at the site - prior to study start.

## 10.6 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to the Clinical Trials Data Bank, http://www.clinicaltrials.gov. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

**Product:** MK-3475

Protocol/Amendment No.:

#### 11.0 APPENDICIES

#### 11.1 ECOG Performance Status

| Grade | Description |
|-------|----------------------------------------------------------------------|
| 0 | Normal activity. Fully active, able to carry on all pre-disease |
| | performance without restriction. |
| | Symptoms, but ambulatory. Restricted in physically strenuous |
| 1 | activity, but ambulatory and able to carry out work of a light or |
| | sedentary nature (e.g., light housework, office work). |
| | In bed <50% of the time. Ambulatory and capable of all self-care, |
| 2 | but unable to carry out any work activities. Up and about more than |
| | 50% of waking hours. |
| 3 | In bed >50% of the time. Capable of only limited self-care, confined |
| 3 | to bed or chair more than 50% of waking hours. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self- |
| 4 | care. Totally confined to bed or chair. |
| 5 | Dead. |

<sup>\*</sup>As published in Am. J. Clin. Oncol.: Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982. The Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair.

# 11.2 Common Terminology Criteria for Adverse Events V4.0 (CTCAE)

The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for adverse event reporting. (http://ctep.cancer.gov/reporting/ctc.html)

#### 11.3 Response Criteria

# 11.3.1 Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Criteria for Evaluating Response in Solid Tumors

RECIST version 1.1\* will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST 1.1, CT is the preferred imaging technique in this study.

\* As published in the European Journal of Cancer:

E.A. Eisenhauer, P. Therasse, J. Bogaerts, L.H. Schwartz, D. Sargent, R. Ford, J. Dancey, S. Arbuck, S. Gwyther, M. Mooney, L. Rubinstein, L. Shankar, L. Dodd, R. Kaplan, D. Lacombe, J. Verweij. New response evaluation criteria in solid tumors: Revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47.

## 11.3.2 Immune related response criteria (irRC)

The irRC [12] will be used in a explorative fashion, and correlation with survival will be assessed. The irRC used is as published in Clinical Cancer Research:

JD Wolchok, A Hoos, S O'Day et al. Guidelines for the Evaluation of Immune Therapy Activity in Solid Tumors: Immune-Related Response Criteria. Clin Cancer Res 2009:15(23)7412-2011.

#### 11.4 Events of Clinical Interest Guidance Document

# PEMBROLIZUMAB PROGRAM

(MK-3475)

# EVENT OF CLINICAL INTEREST GUIDANCE DOCUMENT

Version 5.0



# **REVISION HISTORY LOG**

| Version | Effective<br>Date* | Revision<br>Author | Action |
|---|---|---|---|
| 1 | 08-Aug-2012 | Kevin Gergich | Initial Release of guidance document for MK-3475 |
| 2 | 07-June-2013 | Marty Huber,<br>Kevin Gergich,<br>Holly Brown | Revised title, formerly was "MK-3475 Immune-Related Adverse Event Identification, Evaluation and Management Guidance Document for Investigators" |
| | | | Revised the format of irAE Guidance document, including layout, font, sectioning, etc. for consistency with Sponsor Events of Clinical Interest guidance documents. |
| | | | Modified Categories for irAEs: |
| | | | <ul> <li>Replaced GI with Colitis category.</li> <li>Removed Neurologic category.</li> <li>Added Renal category.</li> </ul> |
| | | | Removed detail in the irAE Guidance document that can be located in the Investigator's Brochure for MK-3475. |
| | | | Removed details regarding non-MK-3475 compounds. |
| | | | Added ECI reporting guidelines. |
| | | | Included a Table Events of Clinical Interest: Immune-Related Adverse Events that includes the key terms. |
| | | | Also placed a pull-out quick-review sheet in the Appendix. |
| | | | 66 |

| : | | | | Updated background, diagnosis and course of treatment details for irAEs. |
|---|---|---|---|---|
| | 3 | 10-Sep-2014 | Marty Huber,<br>Kevin Gergich,<br>Holly Brown | Renamed the document: "Pembrolizumab Program (MK-3475) - Events of Clinical Interest Guidance Document". |
| | | | | Introduced generic name: pembrolizumab (MK-3475) and inserted throughout the document. |
| | | | | Updated Overview – Section 1 |
| | | | | - Clarified the scope of the document and the reporting window for ECIs |
| | | | | - Updated Table 1 with medDRA Preferred Terms for adverse events to correspond with reporting of terms to clinical database, rearranged the order, and updated the reporting criteria. |
| | | | | - Updated the dose modification/discontinuation section to clarify discontinuation and hold terminology. |
| | : | | | Updated Section 2 – ECI Reporting Guidelines |
| | | | | - Clarified that ECIs must be reported to Merck within 24 hours regardless of attribution to study treatment or etiology. |
| | | | | Updated Section 3 |
| | | | | For All Sections, removed the Course of Action for Grade 1 events. |
| | | | | - Section 3.1 Pneumonitis - Moved Pneumonitis to beginning of ECI Section - Updated management guidelines for Grade 2 and Grade 3-4 events |
| | | | | - Section 3.2 Colitis: |

- Updated AE terms and ECI criteria, updated course of action language for clarity
- Section 3.3 Endocrine:
  - Updated ECI criteria and updated course of action language for clarity.
  - Added subsections for hypophysitis, hyperthyroidism and hypothyroidism to clarify management guidelines.
- Section 3.4 Hematologic:
  - New section added.
- Section 3.5: Hepatic:
  - Updated terms and added additional guidance for reporting of DILI ECI; updated course of action for clarity
- Section 3.6 Neurologic:
  - New section added.
- Section 3.7 Ocular:
  - Changed the name of this section from Eye to Ocular
  - Added the term "iritis", updated ECI guidance, and updated course of action language for clarity
- Section 3.8 Renal:
  - Updated section for clarity.
- Section 3.9 Skin:
  - Updated list of terms and added terms for reporting of other skin ECIs; added section 3.9.1: Immediate Evaluation for Potential Skin ECIs
- Section 3.10 Other:

| , | | | | Updated list of terms for clarity; revised course of action for clarity. |
|---|---|---|---|---|
| | | | | - Section 3.11 Infusion Reactions: |
| | | | | - New section added. |
| | | | | - Section 3.12: Follow-up to Resolution: |
| | | | | - New section added. |
| | | | | - Section 4: |
| | | | | - References updated. |
| : | : | | | - Section 5: |
| | | | | - ECI table updated for consistency with Table 1. |
| | | | | - Section 6: Appendix 2 - Past Medical History Related to Dermatologic Event: New section added. |
| | | | | - Section 7: Appendix 3 – Presentation of the Dermatologic Event: New section added. |
| | | | | - Section 8: Appendix 4 – Focused Skin Examination:<br>New section added. |
| | 4 | 04-Dec-2014 | Scot Ebbinghaus,<br>Oswaldo Bracco, | - Table 1 - Updated Endocrine (reported as ECI if ≥ Grade 3 |
| | | | Holly Brown, | or ≥ Grade 2 and resulting in dose modification or use of systemic steroids to treat the AE) Section to include: |
| | | | Kevin Gergich | <ul> <li>Hyperglycemia, if ≥Grade 3 and associated with ketosis or metabolic acidosis (DKA)</li> <li>Created new section in Table 1 – Endocrine</li> </ul> |
| | | | | (reported as ECI) and added: - Type 1 diabetes mellitus (if new onset) - Hepatic: Clarified Transaminase elevations as: |

| | | | <ul> <li>Transaminase elevations (ALT and/or AST)</li> <li>Section 3.2 Colitis <ul> <li>Updated the duration of diarrhea requirments under the Course of Action for Grade 2 and Grade 3</li> </ul> </li> <li>Section 3.3 Endocrine <ul> <li>Clarified Course of Action for hyperthyroidism and hypothyroidism</li> <li>Added Course of Action section for Type 1 diabetes mellitus (if new onset) and ≥ Grade 3 hyperglycemia</li> </ul> </li> <li>Section 5 <ul> <li>Updated Reference Table in Appendix 1</li> </ul> </li> </ul> |
|---|---|---|---|
| 5 | 18-Dec-2014 | Holly Brown | - Section 3.3 Endocrine |
| | | | - Updated the Course of Action for Hypophysitis |
| | | Kevin Gergich | - Merged Grades 2-4 into one course of action |

<sup>\*</sup>Ensure that you are using the most current version of this document.

# TABLE OF CONTENTS

| 1. OVERVIEW | 73 |
|---|---|
| 2. ECI REPORTING GUIDELINES | |
| 3. ECI CATEGORIES AND TERMS | 77 |
| 3.1 Pneumonitis | 78 |
| 3.2 Colitis | 79 |
| 3.3 Endocrine | 81 |
| 3.4 Hematologic | 84 |
| 3.5 Hepatic | 85 |
| 3.6 Neurologic | 87 |
| 3.7 Ocular | 88 |
| 3.8 Renal | 89 |
| 3.9 Skin | 90 |
| 3.9.1. Immediate Evaluation for Potential Skin ECIs | 92 |
| 3.10 Other | 95 |
| 3.11 Infusion Reactions | 97 |
| 3.12 Follow-up to Resolution | 99 |
| 4. REFERENCES | 100 |
| 5. APPENDIX 1 -Events of Clinical Interest (ECI) - Reference Table | 101 |
| 6. APPENDIX 2 – Past Medical History Related to Dermatologic Event | 104 |
| 7. APPENDIX 3 – Presentation of the Dermatologic Event | <del>1</del> 06 |

| 8 | APPENDIX 4 - | - Focused Skin | Examination1 | 04 | ļ |
|---|--------------|----------------|--------------|----|---|
|---|--------------|----------------|--------------|----|---|
## 1. OVERVIEW

The purpose of this document is to provide study sites with guidance on the identification and management of Events of Clinical Interest for the MK-3475 (also known as pembrolizumab) program.

Based on the literature review [1-11], and consideration of mechanism of action of pembrolizumab, potential immune-related adverse events (irAEs) are the primary Event of Clinical Interest (ECI). Immune-related AEs are adverse events associated with the treatment of patients with immunotherapy treatments that appear to be associated with the immune therapy's mechanism of action. Based on these potential irAEs, the sponsor has defined a list of specific adverse event terms (ECIs) that are selected adverse experiences that **must be reported to Merck within 24 hours** from the time the Investigator/physician is aware of such an occurrence, regardless of whether or not the investigator/physician considers the event to be related to study drug(s). In addition, these ECIs require additional detailed information to be collected and entered in the study database. ECIs may be identified through spontaneous patient report and / or upon review of subject data. **Table 1** provides the list of terms and reporting requirements for AEs that must be reported as ECIs for MK-3475 protocols. Of note, the requirement for reporting of ECIs applies to all arms, including comparators, of MK-3475 clinical trials

Given that our current list of events of clinical interest is not comprehensive for all potential immune-related events, it is possible that AEs other than those listed in this document may be observed in patients receiving pembrolizumab. Therefore any Grade 3 or higher event that the investigator/physician considers to be immune-related should be reported as an ECI regardless of whether the specific event term is in Table 1 and reported to Merck within 24 hours from the time the Investigator/physician is aware of such an occurrence. Adverse events that are both an SAE and an ECI should be reported one time as an SAE only, however the event must be appropriately identified as an ECI as well in in the database.

Table 3: Events of Clinical Interest

| Pneumonitis (reported as ECI if ≥ Grade | 2) | |
|---|---|---|
| Acute interstitial pneumonitis | Interstitial lung disease | Pneumonitis |
| Colitis (reported as ECI if ≥ Grade 2 or a | L<br>by grade resulting in dose modification or | use of systemic steroids to treat the AE) |
| Intestinal Obstruction | Colitis | Colitis microscopic |
| Enterocolitis | Enterocolitis hemorrhagic | Gastrointestinal perforation |
| Necrotizing colitis | Diarrhea | |
| Endocrine (reported as ECI if $\geq$ Grade 3 the AE) | or ≥ Grade 2 and resulting in dose mod | ification or use of systemic steroids to treat |
| Adrenal Insufficiency | Hyperthyroidism | Hypophysitis |
| Hypopituitarism | Hypothyroidism | Thyroid disorder |
| Thyroiditis | Hyperglycemia, if ≥Grade 3 and associate | d with ketosis or metabolic acidosis (DKA) |
| Endocrine (reported as ECI) | | |
| Type 1 diabetes mellitus (if new onset) | | |
| Hematologic (reported as ECI if > Crade<br>AE) | 3 or any grade resulting in dose-modific | ation or use of systemic steroids to treat the |
| Autoimmune hemolytic anemia | Aplastic anemia | Thrombotic Thrombocytopenic Purpura (TTP) |
| Idiopathic (or immune) Thrombocytopenia<br>Purpura (ITP) | Disseminated Intravascular Coagulation (DIC) | Haemolytic Uraemic Syndrome (HUS) |
| Any Grade 4 anemia regardless of underlying | g mechanism | , |
| Hereife freported as EQL if $\geq$ Grade $2$ , $\sigma$ | any grade resulting in dose modification or | use of systeme steroids to treat the AND) |
| Hepatitis | Autoimmune hepatitis | Transaminase elevations (ALT and/or AST) |
| Infusion Reservors (reported as BCH for a | ny grado) | |
| Allergic reaction | Anaphylaxis | Cytokine release syndrome |
| Serum sickness | Infusion reactions | Infusion-like reactions |

| Neurologic (reported as ECL for any grade | AND STREET | Property of the Control of the Contr |
|---|---|---|
| Autoimmune neuropathy | Guillain-Barre syndrome | Demyelinating polyneuropathy |
| Myasthenic syndrome | | |
| Ocular (report as ECL if > Grade 2 or any | grade resulting indose modification or i | seroFsystemic steroids to treat the AE) |
| Uveitis | Iritis | |
| Renal (reported as ECL if $\geq$ Grade 2) | | A TOP STORY |
| Nephritis | Nephritis autoimmune | Renal Failure |
| Renal failure acute | Creatinine elevations (report as ECI if modification or use of systemic steroids to | ≥Grade 3 or any grade resulting in dose treat the AE) |
| Skin (reported as FCL for any gredia) | | en er fill gegen folkspille gestellt av det kommen.<br>De skapping folkspille er film fanne gegen folkspille folkspille |
| Dermatitis exfoliative | Erythema multiforme | Stevens-Johnson syndrome |
| Toxic epidermal necrolysis | | |
| Skin (reported as ECLift≥(Grade 3) | | |
| Pruritus | Rash | Rash generalized |
| Rash maculo-papular | | |
| Any rash considered clinically significant in | the physician's judgment | |
| Other (reported as ICH or any goods) | | |
| Myocarditis | Pancreatitis | Pericarditis |
| Any other Grade 3 event which is considered | l immune-related by the physician | |

Each of the events above is described within this guidance document, along with site requirements for reporting these events to the Sponsor. The information collected should be entered into the narrative field(s) of the Adverse Event module in the database (please note, if narrative entry into the database is not available, please use the narrative text box on the 1727/AER Form). If additional Medical History or Concomitant Medications are reported, the Medical History and Concomitant Medication modules in the database must be updated.

In addition, the guidelines include recommendations on the management of these ECIs. These guidelines are intended to be applied when the physician determines the events to be related to pembrolizumab. Note: if after the evaluation the event is determined not to be related, the physician is instructed to follow the ECI reporting guidance but does not need to follow the treatment guidance (below). Therefore, these recommendations should be seen as guidelines and the treating physician should exercise individual clinical judgment based on the patient. For any question of dose modification or other treatment options, the specific language in the protocol should be followed. Any questions pertaining to the collection of this information or management of ECIs should be directed to your local Sponsor contact.

#### **Dose Modification/Discontinuation**

The treatment guidance provides specific direction when to hold and/or discontinue pembrolizumab for each immune related adverse event. Of note, when the guidance states to "discontinue" pembrolizumab this is the permanent discontinuation of treatment with pembrolizumab. "Hold" means to stop treating with pembrolizumab but resumption of treatment may be considered assuming the patient meets the criteria for resumption of treatment.

#### 2. ECI REPORTING GUIDELINES

ECIs are selected non-serious and serious adverse experiences that must be reported to Merck within 24 hours regardless of attribution to study treatment. The AEs listed in this document and any event that meets the ECI criteria (as noted) in Table 1 or in the respective protocol (event term and Grade) must be reported regardless of physician-determined causality with study medication and whether or not considered immune-related by the physician (unless otherwise specified). Physicians/study coordinators/designated site personnel are required to record these experiences as ECIs on the Adverse Experience electronic Case Report Forms (eCRFs) (or on paper) and to provide supplemental information (such as medical history, concomitant medications, investigations, etc.) about the event.

- Please refer to the Data Entry Guidelines (DEGs) for your protocol.
- Please refer to protocol for details on reporting timelines and reporting of Overdose and Drug Induced Liver Injury (DILI).

# 3. ECI CATEGORIES AND TERMS

This section describes the ECI categories and outlines subject management guidelines when an ECI is reported.



## 11.3 3.1 Pneumonitis

The following AE terms, if considered  $\geq$  Grade 2, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Pneumonitis
- Interstitial lung disease
- Acute interstitial pneumonitis

If symptoms indicate possible new or worsening cardiac abnormalities additional testing and/or a cardiology consultation should be considered.

All attempts should be made to rule out other causes such as metastatic disease, bacterial or viral infection. It is important that patients with a suspected diagnosis of pneumonitis be managed as per the guidance below until treatment-related pneumonitis is excluded. Treatment of both a potential infectious etiology and pneumonitis in parallel may be warranted. Management of the treatment of suspected pneumonitis with steroid treatment should not be delayed for a therapeutic trial of antibiotics. If an alternative diagnosis is established, the patient does not require management as below; however the AE should be reported regardless of etiology.

## **Course of Action**

#### Grade 2 events:

- Report as ECI
- Hold pembrolizumab.
- Consider pulmonary consultation with bronchoscopy and biopsy/BAL.
- Consider ID consult
- Conduct an in person evaluation approximately twice per week
- Consider frequent Chest X-ray as part of monitoring
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg/day prednisone or equivalent. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

78



 Second episode of pneumonitis – discontinue pembrolizumab if upon re-challenge the patient develops a second episode of Grade 2 or higher pneumonitis.

#### Grade 3 and 4 events:

- Report as ECI
- Discontinue pembrolizumab.
- Hospitalize patient
- Bronchoscopy with biopsy and/or BAL is recommended.
- Immediately treat with intravenous steroids (methylprednisolone 125 mg IV). When symptoms improve to Grade 1 or less, a high dose oral steroid (prednisone 1 to 2 mg/kg once per day or dexamethasone 4 mg every 4 hours) taper should be started and continued over no less than 4 weeks.
- If IV steroids followed by high dose oral steroids does not reduce initial symptoms within 48 to 72 hours, treat with additional anti-inflammatory measures. Discontinue additional anti-inflammatory measures upon symptom relief and initiate a prolonged steroid taper over 45 to 60 days. If symptoms worsen during steroid reduction, initiate a retapering of steroids starting at a higher dose of 80 or 100 mg followed by a more prolonged taper and administer additional anti-inflammatory measures, as needed
- Add prophylactic antibiotics for opportunistic infections.

## 3.2 Colitis

The following AE terms, if considered ≥ Grade 2 or resulting in dose modification or use of systemic steroids to treat the AE, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Colitis
- Colitis microscopic
- Enterocolitis
- Enterocolitis hemorrhagic
- Gastrointestinal perforation
- Intestinal obstruction
- Necrotizing colitis
- Diarrhea

All attempts should be made to rule out other causes such as metastatic disease, bacterial or parasitic infection, viral gastroenteritis, or the first manifestation of an inflammatory bowel disease by examination for stool leukocytes, stool cultures, a Clostridium difficile titer and endoscopy. However the AE should be reported regardless of etiology.

79



#### **Course of Action**

Grade 2 Diarrhea/Colitis (4-6 stools/day over baseline, dehydration requiring IV fluids < 24 hours, abdominal pain, mucus or blood in stool):

- Report as ECI
- Hold pembrolizumab.
- Symptomatic Treatment
- For Grade 2 diarrhea that persists for greater than 3 days, and for diarrhea with blood and/or mucus.
  - o Consider GI consultation and endoscopy to confirm or rule out colitis
  - o Administer oral corticosteroids (prednisone 1-2 mg/kg QD or equivalent)
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- If symptoms worsen or persist > 3 days treat as Grade 3

Grade 3 Diarrhea/Colitis (or Grade 2 diarrhea that persists for > 1 week):

- Report as ECI
- Hold pembrolizumab.
- Rule out bowel perforation. Imaging with plain films or CT can be useful.
- Recommend consultation with Gastroenterologist and confirmation biopsy with endoscopy.
- Treat with intravenous steroids (methylprednisolone 125 mg) followed by high dose oral steroids (prednisone 1 to 2 mg/kg once per day or dexamethasone 4 mg every 4 hours) When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Taper over 6 to 8 weeks in patients with diffuse and severe ulceration and/or bleeding.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- If IV steroids followed by high dose oral steroids does not reduce initial symptoms within 48 to 72 hours, consider treatment with additional anti-inflammatory measures as described in the literature [5]. Discontinue additional anti-inflammatory measures upon symptom relief and initiate a prolonged steroid taper over 45 to 60 days. If symptoms worsen during steroid reduction, initiate a retapering of steroids starting at a higher dose of 80 or 100 mg followed by a more prolonged taper and administer additional anti-inflammatory measures as needed.

Grade 4 events:

- Report as ECI
- Permanently discontinue pembrolizumab.
- Manage as per Grade 3.

## 3.3 Endocrine

The following AE terms, if considered  $\geq$ Grade 3 or if  $\geq$ Grade 2 and require holding/discontinuation/modification of pembrolizumab dosing, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Adrenal insufficiency
- Hyperthyroidism
- Hypophysitis
- Hypopituitarism
- Hypothyroidism
- Thyroid disorder
- Thyroiditis

All attempts should be made to rule out other causes such as brain metastases, sepsis and/or infection. However the AE should be reported regardless of etiology.

# Hypophysitis or other symptomatic endocrinopathy other than hypo- or hyperthyroidism

## Grade 2-4 events:

- Report as ECI if appropriate
- Hold pembrolizumab
- Rule out infection and sepsis with appropriate cultures and imaging.
- Monitor thyroid function or other hormonal level tests and serum chemistries more frequently until returned to baseline values.
- Pituitary gland imaging should be considered (MRIs with gadolinium and selective cuts of the pituitary can show enlargement or heterogeneity and confirm the diagnosis).
- Treat with prednisone 40 mg p.o. or equivalent per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.



- Hypophysitis with clinically significant adrenal insufficiency and hypotension, dehydration, and electrolyte abnormalities (such as hyponatremia and hyperkalemia) constitutes adrenal crisis.
- Consultation with an endocrinologist may be considered.

#### Hyperthyroidism and Hypothyroidism

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.

Grade 2 hyperthyroidism, Grade 2-4 hypothyroidism events:

- Report as ECI if appropriate (see Table 1)
- Monitor thyroid function or other hormonal level tests and serum chemistries more frequently until returned to baseline values.
- Thyroid hormone and/or steroid replacement therapy to manage adrenal insufficiency.
- Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted.
- In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
- In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- Consultation with an endocrinologist may be considered.

## Grade 3 hyperthyroidism events:

- Report as ECI
- Hold pembrolizumab.
- Rule out infection and sepsis with appropriate cultures and imaging.
- Treat with an initial dose of methylprednisolone 1 to 2 mg/kg intravenously followed by oral prednisone 1 to 2 mg/kg per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 4 hyperthyroidism events:

- Report as ECI
- Discontinue pembrolizumab.
- Manage as per Grade 3



# Type 1 diabetes mellitus (if new onset) and ≥ Grade 3 Hyperglycemia

The following AE terms are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Type I diabetes mellitus (T1DM), if new onset, including diabetic ketoacidosis (DKA)
- Grade 3 or higher hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA).

Immune-mediated diabetes may present as new onset of Type 1 diabetes or an abrupt worsening of pre-existing diabetes associated with laboratorial evidence of beta cell failure. All attempts should be made to rule out other causes such as type 2 diabetes mellitus (T2DM), T2DM decompensation, steroid-induced diabetes, physiologic stress-induced diabetes, or poorly controlled pre-existing diabetes (either T1DM or T2DM), but events meeting the above criteria should be reported as ECIs regardless of etiology. The patients may present with hyperglycemia (abrupt onset or abrupt decompensation) with clinical evidence of diabetic ketoacidosis or laboratory evidence of insulin deficiency, such as ketonuria, laboratory evidence of metabolic acidosis, or low or undetected c-peptide.

#### **Course of Action**

## T1DM should be immediately treated with insulin.

## T1DM or Grade 3-4 Hyperglycemia events:

- Report as ECI if appropriate (see Table 1)
- Hold pembrolizumab for new onset Type 1 diabetes mellitus or Grade 3-4 hyperglycemia associated with evidence of beta cell failure, and resume pembrolizumab when patients are clinically and metabolically stable.
- Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
- Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.
- Consultation with an Endocrinologist is recommended.



- Consider local testing for islet cell antibodies and antibodies to GAD, IA-2, ZnT8, and insulin may be obtained.

## 3.4 Hematologic

The following AE term, if considered Grade ≥3 or requiring dose modification or use of systemic steroids to treat the AE, are considered an ECI and should be reported to the Sponsor within 24 hours of the event:

- Autoimmune hemolytic anemia
- Aplastic anemia
- Disseminated Intravascular Coagulation (DIC)
- Haemolytic Uraemic Syndrome (HUS)
- Idiopathic (or immune) Thrombocytopenia Purpura (ITP)
- Thrombotic Thrombocytopenic Purpura (TTP)
- Any Grade 4 anemia regardless of underlying mechanism

All attempts should be made to rule out other causes such as metastases, sepsis and/or infection. Relevant diagnostic studies such as peripheral blood smear, reticulocyte count, LDH, haptoglobin, bone marrow biopsy or Coomb's test, etc., should be considered to confirm the diagnosis. However the AE should be reported regardless of etiology.

#### **Course of Action**

#### Grade 2 events:

- Report as ECI
- Hold pembrolizumab
- Prednisone 1-2 mg/kg daily may be indicated
- Consider Hematology consultation.
   Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 3 events:

- Report as ECI
- Hematology consultation.
- Hold pembrolizumab Discontinuation should be considered as per specific protocol guidance.

 Treat with methylprednisolone 125 mg iv or prednisone 1-2 mg/kg p.o. (or equivalent) as appropriate

Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 4 events:

- Report as ECI
- Hematology consultation
- Discontinue pembrolizumab for all solid tumor indications; refer to protocol for hematologic malignancies.
- Treat with methylprednisolone 125 mg iv or prednisone 1-2 mg/kg p.o. (or equivalent) as appropriate

# 3.5 Hepatic

The following AE terms, if considered ≥ Grade 2 or greater (or any grade with dose modification or use of systemic steroids to treat the AE), are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Autoimmune hepatitis
- Hepatitis
- Transaminase elevations

All attempts should be made to rule out other causes such as metastatic disease, infection or other hepatic diseases. However the AE should be reported regardless of etiology.

## Drug Induced Liver Injury (DILI)

In addition, the event must be reported as a Drug Induced Liver Injury (DILI) ECI, if the patient meets the laboratory criteria for potential DILI defined as:

- An elevated alanine transaminase (ALT) or aspartate transaminase (AST) lab value that is greater than or equal to three times (3X) the upper limit of normal (ULN) and
- An elevated total bilirubin lab value that is greater than or equal to two times (2X) ULN and

- At the same time, an alkaline phosphatase (ALP) lab value that is less than 2X ULN,
- As a result of within-protocol-specific testing or unscheduled testing.

Note that any hepatic immune ECI meeting DILI criteria should only be reported once as a DILI event.

#### **Course of Action**

#### Grade 2 events:

- Report as ECI
- Hold pembrolizumab when AST or ALT >3.0 to 5.0 times ULN and/or total bilirubin >1.5 to 3.0 times ULN.
- Monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with 0.5-1 mg/kg/day methylprednisolone or oral equivalent and when LFT returns to grade 1 or baseline, taper steroids over at least 1 month, consider prophylactic antibiotics for opportunistic infections, and resume pembrolizumab per protocol
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.
- Permanently discontinue pembrolizumab for patients with liver metastasis who begin treatment with Grade 2 elevation of AST or ALT, and AST or ALT increases ≥50% relative to baseline and lasts >1 week.

#### Grade 3 events:

- Report as ECI
- Discontinue pembrolizumab when AST or ALT >5.0 times ULN and/or total bilirubin >3.0 times ULN.
- Consider appropriate consultation and liver biopsy to establish etiology of hepatic injury, if necessary
- Treat with high-dose intravenous glucocorticosteroids for 24 to 48 hours. When symptoms improve to Grade 1 or less, a steroid taper with dexamethasone 4 mg every 4 hours or prednisone at 1 to 2 mg/kg should be started and continued over no less than 4 weeks.
- If serum transaminase levels do not decrease 48 hours after initiation of systemic steroids, oral mycophenolate mofetil 500 mg every 12 hours may be given. Infliximab is not recommended due to its potential for hepatotoxicity.
- Several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.



## Grade 4 events:

- Report as ECI
- Permanently discontinue pembrolizumab
- Manage patient as per Grade 3 above

## 3.6 Neurologic

The following AE terms, regardless of grade, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Autoimmune neuropathy
- Demyelinating polyneuropathy
- Guillain-Barre syndrome
- Myasthenic syndrome

All attempts should be made to rule out other causes such as metastatic disease, other medications or infectious causes. However the AE should be reported regardless of etiology.

#### **Course of Action**

## Grade 2 events:

- Report as ECI
- Moderate (Grade 2) consider withholding pembrolizumab.
- Consider treatment with prednisone 1-2 mg/kg p.o. daily as appropriate
- Consider Neurology consultation. Consider biopsy for confirmation of diagnosis.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 3 and 4 events:

- Report as ECI
- Discontinue pembrolizumab
  - Obtain neurology consultation. Consider biopsy for confirmation of diagnosis

 Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day. If condition worsens consider IVIG or other immunosuppressive therapies as per local guidelines

When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

#### 3.7 Ocular

The following AE terms, if considered Grade ≥2 or requiring dose modification or use of systemic steroids to treat the AE, is considered an ECI and should be reported to the Sponsor within 24 hours of the event:

- Uveitis
- Iritis

All attempts should be made to rule out other causes such as metastatic disease, infection or other ocular disease (e.g. glaucoma or cataracts). However the AE should be reported regardless of etiology.

#### **Course of Action**

## Grade 2 events:

- Evaluation by an ophthalmologist is strongly recommended.
- Treat with topical steroids such as 1% prednisolone acetate suspension and iridocyclitics.
- Discontinue pembrolizumab as per protocol if symptoms persist despite treatment with topical immunosuppressive therapy.

## Grade 3 events:

- Evaluation by an ophthalmologist is strongly recommended
- Hold pembrolizumab and consider permanent discontinuation as per specific protocol guidance.



- Treat with systemic corticosteroids such as prednisone at a dose of 1 to 2 mg/kg per day. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 4 events:

- Evaluation by an ophthalmologist is strongly recommended
- Permanently discontinue pembrolizumab.
- Treat with corticosteroids as per Grade 3 above

## 3.8 Renal

The following AEs if  $\geq$  Grade 2 are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Nephritis
- Nephritis autoimmune
- Renal failure
- Renal failure acute

Creatinine elevations  $\geq$  Grade 3 or any grade with dose modification or use of systemic steroids to treat the AE.

All attempts should be made to rule out other causes such as obstructive uropathy, progression of disease, or injury due to other chemotherapy agents. A renal consultation is recommended. However the AE should be reported regardless of etiology.

## **Course of Action**

#### Grade 2 events:

- Hold pembrolizumab
- Treatment with prednisone 1-2 mg/kg p.o. daily.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

## Grade 3-4 events:

- Discontinue pembrolizumab
- Renal consultation with consideration of ultrasound and/or biopsy as appropriate
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone IV or equivalent once per day.

When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.

## **3.9 Skin**

## Rash and Pruritus

The following AEs should be considered as ECIs, if  $\geq$  Grade 3 and should be reported to the Sponsor within 24 hours of the event:

- Pruritus
  - Rash
- Rash generalized
- Rash maculo-papular
- In addition to CTCAE Grade 3 rash, any rash that is considered clinically significant, in the physician's judgment, should be treated as an ECI. Clinical significance is left to the physician to determine, and could possibly include rashes such as the following:
  - o rash with a duration >2 weeks; OR
  - o rash that is >10% body surface area; <u>OR</u>
  - o rash that causes significant discomfort not relieved by topical medication or temporary cessation of study drug.

## Other Skin ECIs

The following AEs should <u>always</u> be reported as ECIs, regardless of grade, and should be reported to the Sponsor within 24 hours of the event:

- Dermatitis exfoliative
- Erythema multiforme
- Steven's Johnson syndrome
- Toxic epidermal necrolysis

Please note, the AE should be reported regardless of etiology.

## **Course of Action**

## Grade 2 events:

- Symptomatic treatment should be given such as topical glucocorticosteroids (e.g., betamethasone 0.1% cream or hydrocortisone 1%) or urea-containing creams in combination with oral anti-pruritics (e.g., diphenhydramine HCl or hydroxyzine HCl).
- Treatment with oral steroids is at physician's discretion for Grade 2 events.

#### Grade 3 events:



- Hold pembrolizumab.
- Consider Dermatology Consultation and biopsy for confirmation of diagnosis.
- Treatment with oral steroids is recommended, starting with 1 mg/kg prednisone or equivalent once per day or dexamethasone 4 mg four times orally daily. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks.

#### Grade 4 events:

- Permanently discontinue pembrolizumab.
- Dermatology consultation and consideration of biopsy and clinical dermatology photograph.
- Initiate steroids at 1 to 2 mg/kg prednisone or equivalent. When symptoms improve to Grade
   1 or less, steroid taper should be started and continued over no less than 4 weeks.

#### 3.9.1. Immediate Evaluation for Potential Skin ECIs

## A. Photographs:

Every attempt should be made to get a photograph of the actual ECI skin lesion or rash as soon as possible. Obtain appropriate consent for subject photographs if a consent form addendum is required by your IRB/ERC.

- Take digital photographs of:
  - o the head (to assess mucosal or eye involvement),
  - o the trunk and extremities, and
  - o a close-up of the skin lesion/rash.
- If possible, a ruler should be placed alongside the site of a skin occurrence as a fixed marker of distance.
- The time/date stamp should be set in the 'ON' position for documentation purposes.
- Photographs should be stored with the subject's study records.
- The Sponsor may request copies of photographs. The local study contact (e.g., CRA) will provide guidance to the site, if needed.

## **B. Past Medical History:**



Collect past medical history relevant to the event, using the questions in Appendix 2 (Past Medical History Related to Dermatologic Event) as a guide. Any preexisting conditions not previously reported (e.g., drug allergy) should be entered into the Medical History eCRF.

## C. Presentation of the Event:

Collect information on clinical presentation and potential contributing factors using the questions in Appendix 3 (Presentation of the Dermatologic Event) as a guide. This information should be summarized and entered in narrative format in the AE eCRF. Please use the available free-text fields, such as Signs and Symptoms. Note pertinent negatives where applicable to reflect that the information was collected. Any treatments administered should be entered on the Concomitant Medication eCRF.

# D. Vitals Signs and Standard Laboratory Tests:

Measure vital signs (pulse, sitting BP, oral temperature, and respiratory rate) and record on the Vital Signs eCRF. Perform standard laboratory tests (CBC with manual differential and serum chemistry panel, including LFTs).

## E. Focused Skin Examination:

Perform a focused skin examination using the questions in Appendix 4 (Focused Skin Examination) as a guide. Information should be summarized and entered on the Adverse Experience eCRF as part of the narrative.

## F. Dermatology Consult

Refer the subject to a dermatologist as soon as possible.

- For a "severe rash", the subject must be seen within 1-2 days of reporting the event.
- For clinically significant rash, the subject should be seen within 3-5 days.

The dermatologist should submit a biopsy sample to a certified dermatopathology laboratory or to a pathologist experienced in reviewing skin specimens.

The site should provide the dermatologist with all relevant case history, including copies of clinical photographs and laboratory test results.

94

## 3.10 Other

The following AEs, regardless of grade, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Myocarditis
- Pericarditis
- Pancreatitis
- Any additional Grade 3 or higher event which the physician considers to be immune related

All attempts should be made to rule out other causes. Therapeutic specialists should be consulted as appropriate. However the AE should be reported regardless of etiology.

## **Course of Action**

Grade 2 events or Grade 1 events that do not improve with symptomatic treatment:

- Withhold pembrolizumab.
- Systemic corticosteroids may be indicated.
- Consider biopsy for confirmation of diagnosis.
- If pembrolizumab held and corticosteroid required, manage as per grade 3 below.

## Grade 3 events:

- Hold pembrolizumab
- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day.
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Permanently discontinue for inability to reduce corticosteroid dose to 10 mg or less of prednisone or equivalent per day within 12 weeks. Otherwise, pembrolizumab treatment may be restarted and the dose modified as specified in the protocol

| events: |
|---------|

- Treat with systemic corticosteroids at a dose of 1 to 2 mg/kg prednisone or equivalent once per day.
- Discontinue pembrolizumab

## 3.11 Infusion Reactions

The following AE terms, regardless of grade, are considered ECIs and should be reported to the Sponsor within 24 hours of the event:

- Allergic reaction
- Anaphylaxis
- Cytokine release syndrome
- Serum sickness
- Infusion reactions
- Infusion-like reactions

Please note, the AE should be reported regardless of etiology.

## **Course of Action**

Refer to infusion reaction table in the protocol and below.

# Infusion Reactions

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |
| Grade 2 Requires infusion interruption but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); | Stop Infusion. Additional appropriate medical therapy may include but is not limited to: IV fluids | Subject may be premedicated 1.5h (± 30 minutes) prior to infusion of pembrolizumab with: |
| prophylactic medications indicated for <=24 hrs | Antihistamines NSAIDS | Diphenhydramine 50 mg p.o. (or equivalent dose of antihistamine). |
| | Acetaminophen Narcotics Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. If symptoms resolve within one hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate (e.g. from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the subject should be premedicated for the next scheduled dose. | Acetaminophen 500-1000 mg p.o. (or equivalent dose of antipyretic). |
| | Subjects who develop Grade 2 toxicity despite adequate premedication should be permanently discontinued from further trial treatment administration. | |

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| Grade 3: | Additional appropriate medical therapy may include but is not limited to: | |
| Prolonged (i.e., not rapidly<br>responsive to symptomatic<br>medication and/or brief | IV fluids | |
| interruption of infusion);<br>recurrence of symptoms | Antihistamines | |
| following initial improvement;<br>hospitalization indicated for | NSAIDS | |
| other clinical sequelae (e.g., renal impairment, pulmonary | Acetaminophen | |
| infiltrates) | Narcotics | |
| Grade 4: | Oxygen | |
| Life-threatening; pressor or ventilatory support indicated | Pressors | |
| | Corticosteroids | |
| | Epinephrine | |
| | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | |
| | Hospitalization may be indicated. | |
| | Subject is permanently discontinued from further trial treatment administration. | |

Appropriate resuscitation equipment should be available in the room and a physician readily available during the period of drug administration.

For Further information, please refer to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE) at <a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>

# 3.12 Follow-up to Resolution



Subjects should be followed to resolution. The Adverse Experience eCRF should be updated with information regarding duration and clinical course of the event. Information obtained from the consulting specialist, including diagnosis, should be recorded in the appropriate AE fields. Free-text fields should be used to record narrative information:

- Clinical course of the event
- Course of treatment
- Evidence supporting recovery
- Follow-up to the clinical course

Any treatments administered for the event should also be entered in the Concomitant Medication eCRF.

## 4. REFERENCES

- 1. Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nature Reviews Cancer 2012; 12:252-264.
- Weber JS Practical Management of Immune-Related Adverse Events from Immune Checkpoint Protein Antibodies for the Oncologist. American Society of Clinical Oncology 2012; 1092-9118/10/1-10.
- 3. Weber JS, Ka"hler KC, and Hauschild A. Management of Immune-Related Adverse Events and Kinetics of Response With Ipilimumab. J Clin Oncol 30. 2012. http://jco.ascopubs.org/cgi/doi/10.1200/JCO.2012.41.6750.
- 4. Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, et al. Improved Survival with Ipilimumab in Patients with Metastatic Melanoma. N Engl J Med 363:711-723, 2010.
- Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, et al. Safety, Activity, and Immune Correlates of Anti-PD-1 Antibody in Cancer. N Engl J Med 2012; 366:2443-2454.
- 6. Brahmer JR, Tykodi SS, Chow LQM, Hwu WJ, et al. Safety and Activity of Anti-PD-L1 Antibody in Patients with Advanced Cancer. N Engl J Med 2012; 366:2455-2465.



- 7. Weber J, Thompson JA, Hamid O, et al: A randomized, double-blind, placebo-controlled, phase II study comparing the tolerability and efficacy of ipilimumab administered with or without prophylactic budesonide in patients with unresectable stage III or IV melanoma. Clin Cancer Res 15:5591-5598, 2009.
- 8. Lemech C and Arkenau HT. Novel Treatments for Metastatic Cutaneous Melanoma and the Management of Emergent Toxicities. Clinical Medicine Insights: Oncology 2012:6 53–66.
- 9. Phan GQ, Weber JS, and Sondak VK. CTLA-4 Blockade with Monoclonal Antibodies in Patients with Metastatic Cancer: Surgical Issues. Annals of Surgical Oncology 15(11):3014–3021.
- 10. Bristol-Myers Squibb: YERVOY (ipilimumab): Serious and fatal immune-mediated adverse reactions—YERVOY Risk Evaluation and Mitigation Strategy (REMS). http://www.yervoy.com/hcp/rems.aspx
- 11. Bristol-Myers Squibb: YERVOY (ipilimumab) prescribing information revised March 2011. http://www.accessdata.fda.gov/drugsatfda\_docs/label/2011/125377s0000lbl.pdf

# 5. APPENDIX 1 -EVENTS OF CLINICAL INTEREST (ECI) - REFERENCE TABLE

| Acute interstitial pneumonitis | Interstitial lung disease | Pneumonitis |
|---|---|---|
| िर्वातितः(हरभूकमास्त्री कः छिटा पी ≥ किल्छोट | 2 or may garde assulfing the loss modifies | rfion or use of systemic steroids to treat (life All) |
| ntestinal Obstruction | Colitis | Colitis microscopic |
| Enterocolitis | Enterocolitis hemorrhagic | Gastrointestinal perforation |
| Necrotizing colitis | Diarrhea | |
| Endocrine (reported as ECI if > C | trade 3 of ≥ Greate 2 and resulting in do | sre-modification or use of systemic sterolus-to dr |

| Adrenal Insufficiency | Hyperthyroidism | Hypophysitis |
|---|---|---|
| Hypopituitarism | Hypothyroidism | Thyroid disorder |
| Thyroiditis | Hyperglycemia, if ≥Grade 3 and associate | d with ketosis or metabolic acidosis (DKA) |
| Endocrine (reported as ECI) | | |
| Type 1 diabetes mellitus (if new onset) | | |
| Hematologic (reported as ECI if ≥ Grade AE) | 3 or any grade resulting in dose modifications and the second of the sec | ation or use of systemic steroids to treat the |
| Autoimmune hemolytic anemia | Aplastic anemia | Thrombotic Thrombocytopenic Purpura (TTP) |
| Idiopathic (or immune) Thrombocytopenia<br>Purpura (ITP) | Disseminated Intravascular Coagulation (DIC) | Haemolytic Uraemic Syndrome (HUS) |
| Any Grade 4 anemia regardless of underlyin | g mechanism | |
| Repartic (reparted as ECI if $\geq$ Gradic 2, or | any grade resulting in dose modification or | use of systemic steroids to treat the AE) |
| Hepatitis | Autoimmune hepatitis | Transaminase elevations (ALT and/or AST) |
| Minimision Reactions (reported as ECU for a | nygrado) | |
| Allergic reaction | Anaphylaxis | Cytokine release syndrome |
| Serum sickness | Infusion reactions | Infusion-like reactions |
| Neurologic (reported as ECU for any grad | | |
| Autoimmune neuropathy | Guillain-Barre syndrome | Demyelinating polyneuropathy |
| Myasthenic syndrome | | |
| 1187 To a State British College | | ise of systemic steroids to treatell to AP). |
| Uveitis | Iritis<br> | |
| Rough peppared as 900 if > (Granic 2) | | |
| Nephritis | Nephritis autoimmune | Renal Failure |
| Renal failure acute | Creatinine elevations (report as ECI if modification or use of systemic steroids to | ≥Grade 3 or any grade resulting in dose treat the AE) |



| Skin (reported as ECI for any grade) | <b>在</b> 30 | 。<br>第二十二章 |
|---|---|---|
| Dermatitis exfoliative | Erythema multiforme | Stevens-Johnson syndrome |
| Toxic epidermal necrolysis | | |
| Skin (reported as ECL if ≥ Grade 3) | | |
| Pruritus | Rash | Rash generalized |
| Rash maculo-papular | | |
| Any rash considered clinically significant in | the physician's judgment | |
| Other (reported as ECI for any grade) | | AND THE PROPERTY OF THE PROPER |
| Myocarditis | Pancreatitis | Pericarditis |
| Any other Grade 3 event which is considered | d immune-related by the physician | |

# 6. APPENDIX 2 – PAST MEDICAL HISTORY RELATED TO DERMATOLOGIC EVENT

| Past Medical History: |
|---|
| Any preexisting conditions not previously reported (e.g., drug allergy) should be entered into the Medical History eCRF. |
| 1. Does the subject have any allergies? □ Yes □ No |
| If yes, please obtain the following information: |
| a. Any allergy to drugs (including topical or ophthalmic drugs)? □ Yes □ No |
| List the drug name(s) and describe the type of allergic response (e.g. rash, anaphylaxis, etc): |
| b. Any allergy to external agents, such as laundry detergents, soaps, poison ivy, nickel, etc.? $\hfill \Box$ Yes $\hfill \Box$ No |
| Describe the agent and type of allergic response: |
| c. Any allergy to food? □ Yes □ No |



| | Describe the food and type of allergic response: |
|---|---|
| | d. Any allergy to animals, insects? □ Yes □ No |
| | Describe the allergen and type of allergic response: |
| | e. Any other allergy? □ Yes □ No |
| | Describe the allergen and type of allergic response: |
| 2. Does | the subject have any other history of skin reactions, skin eruptions, or rashes? $\square$ Yes $\square$ No |
| | If so what kind? |
| 3. Has t | the subject ever been treated for a skin condition? □ Yes □ No |
| | If so what kind? |
| 4. Is the | e current finding similar to a past experience? □ Yes □ No |

## 7. APPENDIX 3 – PRESENTATION OF THE DERMATOLOGIC EVENT

## Presentation of the event:

Collect information on clinical presentation and potential contributing factors. Key information should be summarized and entered on the Adverse Experience eCRF. Any treatments administered should be entered on the Concomitant Medication eCRF.

| 1. What is the onset time of the skin reaction, skin eruption, or rash relative to dose of stud | y drug? |
|---|---|
| 2. Has the subject contacted any known allergens? □ Yes □ No | |
| If so what kind? | |
| 3. Has the subject contacted new, special, or unusual substances (e.g., new laundry detergent personal care product, poison ivy, etc.)? $\Box$ Yes $\Box$ No | ts, soap, |
| If so what kind? | |
| 4. Has the subject taken any other medication (over the counter, prescription, vitami supplement)? □ Yes □ No | ns, and |
| If so what kind? | |
| 5. Has the subject consumed unaccustomed, special or unusual foods? □ Yes □ No | |
| If so what kind? | |



| 6. Does the subject have or had in the last few days any illness? □ Yes □ No |
|---|
| If so what kind? |
| 7. Has the subject come into contact with any family or house members who are ill? □ Yes □ No |
| If so who and what? |
| 8. Has the subject recently been near children who have a skin reaction, skin eruption, or rash (e.g. <i>Molluscum Contagiosum</i> )? □ Yes □ No |

| 9. Has the subject had recent sun exposure? □ Yes □ No |
|---|
| 10. For the current rash, have there been any systemic clinical signs? □ Yes □ No |
| If so what kind? |
| i. Anaphylaxis? □ Yes □ No |
| ii. Signs of hypotension? □ Yes □ No |
| iii. Signs of dyspnea? □ Yes □ No iv. Fever, night sweats, chills? □ Yes □ No |
| 11. For the current rash, has the subject needed subcutaneous epinephrine or other systemic catecholamine therapy? Yes No If so what kind? |
| 12. For the current rash, has the subject used any other medication, such as inhaled bronchodilators antihistaminic medication, topical corticosteroid, and/or systemic corticosteroid? □ Yes □ No |
| List medication(s) and dose(s): |
| 13. Is the rash pruritic (itchy)? □ Yes □ No |



# APPENDIX 4 – FOCUSED SKIN EXAMINATION

| Focused S | kin Examin | ation: | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Key inforn | nation should | l be sur | nmarized an | d ente | ered on | the Adverse | Exper | ience eCRF. | | |
| Primary Skin Lesions Description | | | | | | | | | | |
| Color: | | | | <del></del> . | | | | _ | | |
| General de | scription: | | | | | | | | | |
| | | | | | | | | 1 | | |
| | ne distributio | | | | | | | | | |
| | | | | | | | | . <del></del> | | |
| | reaction, | | eruption, | | | | | continuing | to | spread? |
| Any | associated | | signs | | on | | physical | | examination? | |

#### 12.1 REFERENCES:

- 1. Lee HY, Chay WY, Tang MB et al. Melanoma: differences between Asian and Caucasian patients. Ann Acad Med Singapore 2012; 41: 17-20.
- 2. Green A, McCredie M, MacKie R et al. A case-control study of melanomas of the soles and palms (Australia and Scotland). Cancer Causes Control 1999; 10: 21-25.
- 3. Jung HJ, Kweon SS, Lee JB et al. A clinicopathologic analysis of 177 acral melanomas in Koreans: relevance of spreading pattern and physical stress. JAMA Dermatol 2013; 149: 1281-1288.
- 4. Curtin JA, Fridlyand J, Kageshita T et al. Distinct sets of genetic alterations in melanoma. N Engl J Med 2005; 353: 2135-2147.
- 5. Curtin JA, Busam K, Pinkel D, Bastian BC. Somatic activation of KIT in distinct subtypes of melanoma. J Clin Oncol 2006; 24: 4340-4346.
- 6. Furney SJ, Turajlic S, Fenwick K et al. Genomic characterisation of acral melanoma cell lines. Pigment Cell Melanoma Res 2012; 25: 488-492.
- 7. Furney SJ, Turajlic S, Stamp G et al. The mutational burden of acral melanoma revealed by whole-genome sequencing and comparative analysis. Pigment Cell Melanoma Res 2014; 27: 835-838.
- 8. Poole RM. Pembrolizumab: first global approval. Drugs 2014; 74: 1973-1981.
- 9. Weber J. Immunotherapy for melanoma. Curr Opin Oncol 2011; 23: 163-169.
- 10. Robert C, Ribas A, Wolchok JD et al. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet 2014; 384: 1109-1117.
- 11. Eisenhauer EA, Therasse P, Bogaerts J et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer 2009; 45: 228-247.
- 12. Wolchok JD, Hoos A, O'Day S et al. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res 2009; 15: 7412-7420.